CLINICAL TRIAL: NCT00526474
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of SCH 530348 in Addition to Standard of Care in Subjects With a History of Atherosclerotic Disease: Thrombin Receptor Antagonist in Secondary Prevention of Atherothrombotic Ischemic Events (TRA 2°P - TIMI 50)
Brief Title: Trial to Assess the Effects of Vorapaxar (SCH 530348; MK-5348) in Preventing Heart Attack and Stroke in Patients With Atherosclerosis (TRA 2°P - TIMI 50) (P04737)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: The TIMI Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: P04737; TRA 2°P - TIMI 50; 2006-002942-12; MK-5348-015 (Other: Merck Study Number)
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Results first posted 2014-06-18 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2018-08

CONDITIONS: Atherosclerosis; Ischemia; Myocardial Infarction; Cerebrovascular Accident; Peripheral Arterial Disease
MeSH Terms: conditions — Atherosclerosis; Ischemia; Myocardial Infarction; Stroke; Peripheral Arterial Disease | interventions — vorapaxar

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 1 placebo tablet, orally, daily for at least 1 year in addition to current treatment of atherosclerotic disease, which will be continued to be administered as per current standard of care.
  Interventions: Drug: Placebo
- Vorapaxar (Experimental): one 2.5 mg tablet daily, orally, for at least 1 year in addition to current treatment of atherosclerotic disease, which will be continued to be administered as per current standard of care.
  Interventions: Drug: Vorapaxar

INTERVENTIONS:
Drug: Vorapaxar — 2.5-mg tablet daily for at least 1 year
  Arms: Vorapaxar
Drug: Placebo — matching tablet daily for at least 1 year
  Arms: Placebo

SUMMARY:
The study is designed to determine whether vorapaxar, when added to the existing standard of care (SOC) for preventing heart attack and stroke (eg, aspirin, clopidogrel) in participants with a known history of atherosclerosis, will yield additional benefit over the existing standard of care without vorapaxar in preventing heart attack and stroke.

The study is also designed to assess risk of bleeding with vorapaxar added to the standard of care versus the standard of care alone.

ELIGIBILITY:
Inclusion Criteria:

Men and women at least 18 years old with evidence or a history of atherosclerosis involving the coronary, cerebral, or peripheral vascular systems by one or more of the following:

* history of myocardial infarction (heart attack)
* history of ischemic stroke (stroke due to a blocked artery)
* history of peripheral arterial disease

Exclusion Criteria:

* history of intracranial hemorrhage or of central nervous system (CNS) surgery, tumor, or aneurysm
* any bleeding disorder or abnormality
* sustained severe hypertension or valvular heart disease
* current or recent platelet count <100,000 mm^3
* planned or ongoing treatment with a blood thinning medication
* pregnancy
* any significant medical or physiological condition or abnormality that could put the subject at increased risk or limit the subject's ability to participate for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26449 (Actual)
Dates: Start 2007-09-01 (Actual); Primary Completion 2011-12-01 (Actual); Study Completion 2011-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730
- [Derived] Berg DD, Freedman BL, Bonaca MP, Jarolim P, Scirica BM, Goodrich EL, Sabatine MS, Morrow DA. Cardiovascular Biomarkers and Heart Failure Risk in Stable Patients With Atherothrombotic Disease: A Nested Biomarker Study From TRA 2 degrees P-TIMI 50. J Am Heart Assoc. 2021 May 4;10(9):e018673. doi: 10.1161/JAHA.120.018673. Epub 2021 Apr 22. PMID 33884889
- [Derived] Qamar A, Morrow DA, Creager MA, Scirica BM, Olin JW, Beckman JA, Murphy SA, Bonaca MP. Effect of vorapaxar on cardiovascular and limb outcomes in patients with peripheral artery disease with and without coronary artery disease: Analysis from the TRA 2 degrees P-TIMI 50 trial. Vasc Med. 2020 Apr;25(2):124-132. doi: 10.1177/1358863X19892690. Epub 2020 Jan 30. PMID 32000630
- [Derived] Xu H, Bonaca MP, Goodrich E, Scirica BM, Morrow DA. Efficacy and safety of vorapaxar for secondary prevention in low body weight in patients with atherosclerosis: analyses from the TRA 2 degrees P-TIMI 50 Trial. Eur Heart J Acute Cardiovasc Care. 2021 Apr 8;10(2):190-199. doi: 10.1177/2048872619883354. Epub 2019 Oct 23. PMID 31642690
- [Derived] Bonaca MP, Creager MA, Olin J, Scirica BM, Gilchrist IC Jr, Murphy SA, Goodrich EL, Braunwald E, Morrow DA. Peripheral Revascularization in Patients With Peripheral Artery Disease With Vorapaxar: Insights From the TRA 2 degrees P-TIMI 50 Trial. JACC Cardiovasc Interv. 2016 Oct 24;9(20):2157-2164. doi: 10.1016/j.jcin.2016.07.034. PMID 27765312
- [Derived] Bohula EA, Bonaca MP, Braunwald E, Aylward PE, Corbalan R, De Ferrari GM, He P, Lewis BS, Merlini PA, Murphy SA, Sabatine MS, Scirica BM, Morrow DA. Atherothrombotic Risk Stratification and the Efficacy and Safety of Vorapaxar in Patients With Stable Ischemic Heart Disease and Previous Myocardial Infarction. Circulation. 2016 Jul 26;134(4):304-13. doi: 10.1161/CIRCULATIONAHA.115.019861. PMID 27440003
- [Derived] Kidd SK, Bonaca MP, Braunwald E, De Ferrari GM, Lewis BS, Merlini PA, Murphy SA, Scirica BM, White HD, Morrow DA. Universal Classification System Type of Incident Myocardial Infarction in Patients With Stable Atherosclerosis: Observations From Thrombin Receptor Antagonist in Secondary Prevention of Atherothrombotic Ischemic Events (TRA 2 degrees P)-TIMI 50. J Am Heart Assoc. 2016 Jul 18;5(7):e003237. doi: 10.1161/JAHA.116.003237. PMID 27431644
- [Derived] Berg DD, Bonaca MP, Braunwald E, Corbalan R, Goto S, Kiss RG, Murphy SA, Scirica BM, Spinar J, Morrow DA. Outcomes in Stable Patients With Previous Atherothrombotic Events Receiving Vorapaxar Who Experience a New Acute Coronary Event (from TRA2 degrees P-TIMI 50). Am J Cardiol. 2016 Apr 1;117(7):1055-8. doi: 10.1016/j.amjcard.2015.12.052. Epub 2016 Jan 14. PMID 26876014
- [Derived] Bonaca MP, Gutierrez JA, Creager MA, Scirica BM, Olin J, Murphy SA, Braunwald E, Morrow DA. Acute Limb Ischemia and Outcomes With Vorapaxar in Patients With Peripheral Artery Disease: Results From the Trial to Assess the Effects of Vorapaxar in Preventing Heart Attack and Stroke in Patients With Atherosclerosis-Thrombolysis in Myocardial Infarction 50 (TRA2 degrees P-TIMI 50). Circulation. 2016 Mar 8;133(10):997-1005. doi: 10.1161/CIRCULATIONAHA.115.019355. Epub 2016 Jan 29. PMID 26826179
- [Derived] Bohula EA, Aylward PE, Bonaca MP, Corbalan RL, Kiss RG, Murphy SA, Scirica BM, White H, Braunwald E, Morrow DA. Efficacy and Safety of Vorapaxar With and Without a Thienopyridine for Secondary Prevention in Patients With Previous Myocardial Infarction and No History of Stroke or Transient Ischemic Attack: Results from TRA 2 degrees P-TIMI 50. Circulation. 2015 Nov 17;132(20):1871-9. doi: 10.1161/CIRCULATIONAHA.114.015042. Epub 2015 Sep 3. PMID 26338971
- [Derived] Magnani G, Bonaca MP, Braunwald E, Dalby AJ, Fox KA, Murphy SA, Nicolau JC, Oude Ophuis T, Scirica BM, Spinar J, Theroux P, Morrow DA. Efficacy and safety of vorapaxar as approved for clinical use in the United States. J Am Heart Assoc. 2015 Mar 19;4(3):e001505. doi: 10.1161/JAHA.114.001505. PMID 25792124
- [Derived] Cavender MA, Scirica BM, Bonaca MP, Angiolillo DJ, Dalby AJ, Dellborg M, Morais J, Murphy SA, Ophuis TO, Tendera M, Braunwald E, Morrow DA. Vorapaxar in patients with diabetes mellitus and previous myocardial infarction: findings from the thrombin receptor antagonist in secondary prevention of atherothrombotic ischemic events-TIMI 50 trial. Circulation. 2015 Mar 24;131(12):1047-53. doi: 10.1161/CIRCULATIONAHA.114.013774. Epub 2015 Feb 13. PMID 25681464
- [Derived] Bonaca MP, Scirica BM, Braunwald E, Wiviott SD, Goto S, Nilsen DW, Bonarjee V, Murphy SA, Morrow DA. New ischemic stroke and outcomes with vorapaxar versus placebo: results from the TRA 2 degrees P-TIMI 50 trial. J Am Coll Cardiol. 2014 Dec 9;64(22):2318-26. doi: 10.1016/j.jacc.2014.07.997. Epub 2014 Dec 1. PMID 25465417
- [Derived] Bonaca MP, Scirica BM, Braunwald E, Wiviott SD, O'Donoghue ML, Murphy SA, Morrow DA. Coronary stent thrombosis with vorapaxar versus placebo: results from the TRA 2 degrees P-TIMI 50 trial. J Am Coll Cardiol. 2014 Dec 9;64(22):2309-17. doi: 10.1016/j.jacc.2014.09.037. Epub 2014 Dec 1. PMID 25465416
- [Derived] Bonaca MP, Scirica BM, Creager MA, Olin J, Bounameaux H, Dellborg M, Lamp JM, Murphy SA, Braunwald E, Morrow DA. Vorapaxar in patients with peripheral artery disease: results from TRA2degreesP-TIMI 50. Circulation. 2013 Apr 9;127(14):1522-9, 1529e1-6. doi: 10.1161/CIRCULATIONAHA.112.000679. Epub 2013 Mar 15. PMID 23501976
- [Derived] Morrow DA, Alberts MJ, Mohr JP, Ameriso SF, Bonaca MP, Goto S, Hankey GJ, Murphy SA, Scirica BM, Braunwald E; Thrombin Receptor Antagonist in Secondary Prevention of Atherothrombotic Ischemic Events-TIMI 50 Steering Committee and Investigators. Efficacy and safety of vorapaxar in patients with prior ischemic stroke. Stroke. 2013 Mar;44(3):691-8. doi: 10.1161/STROKEAHA.111.000433. Epub 2013 Feb 8. PMID 23396280
- [Derived] Scirica BM, Bonaca MP, Braunwald E, De Ferrari GM, Isaza D, Lewis BS, Mehrhof F, Merlini PA, Murphy SA, Sabatine MS, Tendera M, Van de Werf F, Wilcox R, Morrow DA; TRA 2 degrees P-TIMI 50 Steering Committee Investigators. Vorapaxar for secondary prevention of thrombotic events for patients with previous myocardial infarction: a prespecified subgroup analysis of the TRA 2 degrees P-TIMI 50 trial. Lancet. 2012 Oct 13;380(9850):1317-24. doi: 10.1016/S0140-6736(12)61269-0. Epub 2012 Aug 26. PMID 22932716
- [Derived] Morrow DA, Braunwald E, Bonaca MP, Ameriso SF, Dalby AJ, Fish MP, Fox KA, Lipka LJ, Liu X, Nicolau JC, Ophuis AJ, Paolasso E, Scirica BM, Spinar J, Theroux P, Wiviott SD, Strony J, Murphy SA; TRA 2P-TIMI 50 Steering Committee and Investigators. Vorapaxar in the secondary prevention of atherothrombotic events. N Engl J Med. 2012 Apr 12;366(15):1404-13. doi: 10.1056/NEJMoa1200933. Epub 2012 Mar 24. PMID 22443427
- [Derived] Morrow DA, Scirica BM, Fox KA, Berman G, Strony J, Veltri E, Bonaca MP, Fish P, McCabe CH, Braunwald E; TRA 2(o)P-TIMI 50 Investigators. Evaluation of a novel antiplatelet agent for secondary prevention in patients with a history of atherosclerotic disease: design and rationale for the Thrombin-Receptor Antagonist in Secondary Prevention of Atherothrombotic Ischemic Events (TRA 2 degrees P)-TIMI 50 trial. Am Heart J. 2009 Sep;158(3):335-341.e3. doi: 10.1016/j.ahj.2009.06.027. PMID 19699854
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=P04737&kw=P04737&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prior to planned study completion, the Data Safety Monitoring Board (DSMB) recommended discontinuation of study drug in all participants with a pre- or post-randomization history of stroke. A total of 4510 participants had study medication stopped, however these participants were included in the overall population for efficacy and safety analyses.
Pre-assignment Details: The Intent to Treat (ITT) Population, defined as all enrolled participants who were randomly assigned to a treatment group.
Period: Overall Study
Arm/Group | Placebo | Vorapaxar
Started | 13224 | 13225
Received Study Drug | 13166 | 13186
Completed | 12932 | 12953
Not Completed | 292 | 272

BASELINE CHARACTERISTICS:
Population: The Intent to Treat (ITT) Population, defined as all enrolled participants who were randomly assigned to a treatment group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vorapaxar | Total
Number analyzed (Participants) | 13224 | 13225 | 26449
Age, Customized [Number; unit: Participants]
  <65 years | 8273 | 8188 | 16461
  65-<75 years | 3445 | 3523 | 6968
  >=75 years | 1506 | 1514 | 3020
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3172 | 3154 | 6326
  Male | 10052 | 10071 | 20123

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced Cardiovascular (CV) Death, Myocardial Infarction (MI), Stroke, or Urgent Coronary Revascularization (UCR) Within 3 Years From Randomization
Description: The time (in days) from study start to the first occurrence of any of the following clinical outcomes was recorded: CV death, MI, stroke, or UCR. A Clinical Endpoints Committee (CEC) reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). If a participant had a fatal event that was not part of a specific endpoint for analysis, they were censored at the time of death. The Kaplan-Meier estimate reports the percentage of participants who experienced CV death, MI, stroke, or UCR within 3 years from randomization.
Time Frame: up to 3 years
Population: Intent to Treat (ITT) Population, defined as all participants who were randomly assigned to a treatment arm.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 13224 | 13225
Percentage of Participants | 12.4 | 11.2
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p = 0.001, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.88, 95% CI 2-sided [0.82 to 0.95] — Hazard ratio calculated by dividing the Kaplan-Meier (KM) Estimate for vorapaxar by the KM Estimate for Placebo and correcting for covariates. A hazard ratio <1 would indicate a lower hazard associated with vorapaxar relative to placebo

2. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced CV Death, MI, or Stroke Within 3 Years From Randomization
Description: The time (in days) from study start to the first occurrence of any of the following clinical outcomes was recorded: CV death, MI, or stroke. A CEC reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). If a participant had a fatal event that was not part of a specific endpoint for analysis, they were censored at the time of death. The Kaplan-Meier estimate reports the percentage of participants who experienced CV death, MI, or stroke within 3 years from randomization.
Time Frame: up to 3 years
Population: ITT Population, defined as all participants who were randomly assigned to a treatment arm.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 13224 | 13225
Percentage of Participants | 10.5 | 9.3
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p < 0.001, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.87, 95% CI 2-sided [0.80 to 0.94] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Met Global Utilization of Streptokinase and Tissue Plasminogen Activator for Occluded Arteries (GUSTO) Moderate or Severe Bleeding Criteria Within 3 Years From Randomization
Description: Adverse events were categorized as "bleeding events" if the intensity, frequency, or type of the event was other or more than would be normally expected in the given situation (eg, mild nosebleed in a person who does not normally have nosebleeds, greater bruising than expected for a given injury, greater volume of blood loss than expected for a given procedure). The investigator graded the intensity of bleeding events according to the GUSTO cooperative group criteria as follows: Mild , Moderate or Severe and the grading was adjudicated by the CEC. The Kaplan-Meier estimate reports the percentage of participants who experienced GUSTO moderate or severe bleeding within 3 years from randomization.
Time Frame: up to 3 years
Population: As Treated Population, which included all participants who received at least 1 dose of study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 13166 | 13186
Percentage of Participants | 2.9 | 4.2
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p < 0.001, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 1.51, 95% CI 2-sided [1.31 to 1.74] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced Clinically Significant Bleeding Within 3 Years From Randomization
Description: Adverse events were categorized as "bleeding events" if the intensity, frequency, or type of the event was other or more than would be normally expected in the given situation (eg, mild nosebleed in a person who does not normally have nosebleeds, greater bruising than expected for a given injury, greater volume of blood loss than expected for a given procedure). The investigator graded the intensity of bleeding events according to the Thrombolysis in Myocardial Infarction (TIMI) Study Group criteria as major, minor or other. "Clinically Significant Bleeding" was defined as the composite of TIMI Major bleeding, TIMI Minor bleeding, or bleeding that required unplanned medical or surgical treatment or unplanned laboratory evaluation even if it did not meet the criteria for TIMI major or minor bleeding. The Kaplan-Meier estimate reports the percentage of participants who experienced clinically significant bleeding within 3 years from randomization.
Time Frame: up to 3 years
Population: As Treated Population, which included all participants who received at least 1 dose of study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 13166 | 13186
Percentage of Participants | 11.3 | 15.4
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p < 0.001, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 1.41, 95% CI 2-sided [1.31 to 1.51] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced Death From Any Cause, MI, Stroke, or UCR Within 3 Years From Randomization
Description: The time (in days) from study start to the occurrence of any of the following clinical outcomes was recorded: death from any cause, MI, stroke, or UCR. A CEC reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). The Kaplan-Meier estimate reports the percentage of participants who experienced death from any cause, MI, stroke, or UCR within 3 years from randomization.
Time Frame: up to 3 years
Population: ITT Population, defined as all participants who were randomly assigned to a treatment arm.
Measure: Number; unit: Perentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 13224 | 13225
Perentage of Participants | 14.2 | 13.2
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p = 0.009, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.91, 95% CI 2-sided [0.85 to 0.98] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced CV Death or an MI Within 3 Years From Randomization
Description: The time (in days) from study start to the occurrence of CV death or MI. A CEC reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). If a participant had a fatal event that was not part of a specific endpoint for analysis, they were censored at the time of death. The Kaplan-Meier estimate reports the percentage of participants who experienced CV death or MI within 3 years from randomization.
Time Frame: up to 3 years
Population: ITT Population, defined as all participants who were randomly assigned to a treatment arm.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 13224 | 13225
Percentage of Participants | 8.2 | 7.3
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p = 0.002, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.86, 95% CI 2-sided [0.78 to 0.94] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced CV Death, MI, Stroke, UCR, or Urgent Hospitalization for Vascular Cause of Ischemic Nature (UH-VCIN) Within 3 Years From Randomization
Description: The time (in days) from study start to the first occurrence of any of the following clinical outcomes was recorded: CV death, MI, stroke, UCR or UH-VCIN. A CEC reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). If a participant had a fatal event that was not part of a specific endpoint for analysis, they were censored at the time of death. The Kaplan-Meier estimate reports the percentage of participants who experienced CV death, MI, stroke, UCR, or UH-VCIN within 3 years from randomization.
Time Frame: up to 3 years
Population: ITT Population, defined as all participants who were randomly assigned to a treatment arm.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 13224 | 13225
Percentage of Participants | 14.7 | 13.1
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p < 0.001, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.87, 95% CI 2-sided [0.81 to 0.93] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Died From Any Cause, or Experienced an MI, Stroke, or Any Revascularization Within 3 Years From Randomization
Description: The time (in days) from study start to death from any cause or the first occurrence of any of the following clinical outcomes was recorded: MI, stroke, or any revascularization procedure . A CEC reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). The Kaplan-Meier estimate reports the percentage of participants who died from any cause, or experienced an MI, stroke, or any revascularization within 3 years from randomization.
Time Frame: up to 3 years
Population: ITT Population, defined as all participants who were randomly assigned to a treatment arm.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 13224 | 13225
Percentage of Participants | 22.6 | 20.7
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p = 0.001, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.91, 95% CI 2-sided [0.86 to 0.96] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced CV Death, MI, Stroke, Any Revascularization, or UH-VCIN Within 3 Years From Randomization
Description: The time (in days) from study start to the first occurrence of any of the following clinical outcomes was recorded: CV death, MI, stroke, any revascularization, or UH-VCIN. A CEC reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). If a participant had a fatal event that was not part of a specific endpoint for analysis, they were censored at the time of death. The Kaplan-Meier estimate reports the percentage of participants who experienced CV death, MI, stroke, any revascularization procedure, or UH-VCIN within 3 years from randomization.
Time Frame: up to 3 years
Population: ITT Population, defined as all participants who were randomly assigned to a treatment arm.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 13224 | 13225
Percentage of Participants | 22.1 | 19.9
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p < 0.001, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.90, 95% CI 2-sided [0.85 to 0.95] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced CV Death Within 3 Years From Randomization
Description: The time (in days) from study start to CV death (if reported) was recorded. A CEC reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). If a participant had a fatal event that was not part of a specific endpoint for analysis, they were censored at the time of death. The Kaplan-Meier estimate reports the percentage of participants who experienced CV death within 3 years from randomization.
Time Frame: up to 3 years
Population: ITT Population, defined as all participants who were randomly assigned to a treatment arm.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 13224 | 13225
Percentage of Participants | 3.0 | 2.7
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p = 0.151, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.89, 95% CI 2-sided [0.76 to 1.04] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced an MI Within 3 Years From Randomization
Description: The time (in days) from study start to the first occurrence of an MI was recorded. A CEC reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). If a participant had a fatal event that was not part of a specific endpoint for analysis, they were censored at the time of death. The Kaplan-Meier estimate reports the percentage of participants who experienced an MI within 3 years from randomization.
Time Frame: up to 3 years
Population: ITT Population, defined as all participants who were randomly assigned to a treatment arm.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 13224 | 13225
Percentage of Participants | 6.1 | 5.2
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p = 0.001, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.83, 95% CI 2-sided [0.74 to 0.93] — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced UCR Within 3 Years From Randomization
Description: The time (in days) from study start to the first occurrence of UCR was recorded. A CEC reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). If a participant had a fatal event that was not part of a specific endpoint for analysis, they were censored at the time of death. The Kaplan-Meier estimate reports the percentage of participants who experienced UCR within 3 years from randomization.
Time Frame: up to 3 years
Population: ITT Population, defined as all participants who were randomly assigned to a treatment arm.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 13224 | 13225
Percentage of Participants | 2.6 | 2.5
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p = 0.108, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.88, 95% CI 2-sided [0.75 to 1.03] — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced a Stroke Within 3 Years From Randomization
Description: The time (in days) from study start to first experience of a stroke was recorded. A CEC reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). If a participant had a fatal event that was not part of a specific endpoint for analysis, they were censored at the time of death. The Kaplan-Meier estimate reports the percentage of participants who experienced a stroke within 3 years from randomization.
Time Frame: up to 3 years
Population: ITT Population, defined as all participants who were randomly assigned to a treatment arm.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 13224 | 13225
Percentage of Participants | 2.8 | 2.8
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p = 0.733, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.97, 95% CI 2-sided [0.83 to 1.14] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Died From Any Cause Within 3 Years From Randomization
Description: The time (in days) from study start to death from any cause was recorded. A CEC reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). The Kaplan-Meier estimate reports the percentage of participants who died from any cause within 3 years from randomization.
Time Frame: up to 3 years
Population: ITT Population, defined as all participants who were randomly assigned to a treatment arm.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 13224 | 13225
Percentage of Participants | 5.3 | 5.0
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p = 0.411, Cox Proportional Hazards Regression; Cox Proportional Hazard = 0.95, 95% CI 2-sided [0.85 to 1.07] — [estimate comment as in outcome 1, analysis 1]

15. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Had a UH-VCIN Within 3 Years From Randomization
Description: The time (in days) from study start to the first occurrence of an UH-VCIN was recorded. A CEC reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). If a participant had a fatal event that was not part of a specific endpoint for analysis, they were censored at the time of death. The Kaplan-Meier estimate reports the percentage of participants who had a UH-VCIN within 3 years from randomization.
Time Frame: up to 3 years
Population: ITT Population, defined as all participants who were randomly assigned to a treatment arm.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 13224 | 13225
Percentage of Participants | 5.5 | 4.7
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p = 0.001, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.83, 95% CI 2-sided [0.74 to 0.93] — [estimate comment as in outcome 1, analysis 1]

16. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Had Any Revascularization Performed Within 3 Years From Randomization
Description: The time (in days) from study start to the first occurrence of a revascularization was recorded. A CEC reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). If a participant had a fatal event that was not part of a specific endpoint for analysis, they were censored at the time of death. The Kaplan-Meier estimate reports the percentage of participants who had any revascularization performed within 3 years from randomization.
Time Frame: up to 3 years
Population: ITT Population, defined as all participants who were randomly assigned to a treatment arm.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 13224 | 13225
Percentage of Participants | 15.5 | 13.6
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p < 0.001, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.89, 95% CI 2-sided [0.83 to 0.95] — [estimate comment as in outcome 1, analysis 1]

17. Post Hoc Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced CV Death, MI, Stroke, or UCR Within 3 Years From Randomization
Description: The time (in days) from study start to the first occurrence of any of the following clinical outcomes was recorded: CV death, MI, stroke, or UCR. A CEC reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). If a participant had a fatal event that was not part of a specific endpoint for analysis, they were censored at the time of death. The Kaplan-Meier estimate reports the percentage of participants who experienced CV death, MI, stroke, or UCR within 3 years from randomization.
Time Frame: up to 3 years
Population: Intended Label Population: all enrolled participants with coronary arterial disease (CAD) or peripheral arterial disease (PAD) and no history of a stroke or transient ischemic attack (TIA)
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 10090 | 10080
Percentage of Participants | 11.8 | 10.1
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p < 0.001, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.83, 95% CI 2-sided [0.76 to 0.90] — [estimate comment as in outcome 1, analysis 1]

18. Post Hoc Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced CV Death, MI, or Stroke Within 3 Years From Randomization
Description: as for outcome 2
Time Frame: up to 3 years
Population: Intended Label Population: all enrolled participants with CAD or PAD and no history of a stroke or TIA
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 10090 | 10080
Percentage of Participants | 9.5 | 7.9
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p < 0.001, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.80, 95% CI 2-sided [0.73 to 0.89] — [estimate comment as in outcome 1, analysis 1]

19. Post Hoc Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Met GUSTO Moderate or Severe Bleeding Criteria Within 3 Years From Randomization
Description: as for outcome 3
Time Frame: up to 3 years
Population: Intended Label Safety Population: all enrolled participants with CAD or PAD and no history of a stroke or TIA who received at least 1 dose of study drug
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 10049 | 10059
Percentage of Participants | 2.7 | 3.8
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p < 0.001, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 1.45, 95% CI 2-sided [1.23 to 1.71] — [estimate comment as in outcome 1, analysis 1]

20. Post Hoc Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced Clinically Significant Bleeding Within 3 Years From Randomization
Description: Adverse events were categorized as "bleeding events" if the intensity, frequency, or type of the event was other or more than would be normally expected in the given situation (eg, mild nosebleed in a person who does not normally have nosebleeds, greater bruising than expected for a given injury, greater volume of blood loss than expected for a given procedure). The investigator graded the intensity of bleeding events according to the TIMI Study Group criteria as major, minor or other. "Clinically Significant Bleeding" was defined as the composite of TIMI Major bleeding, TIMI Minor bleeding, or bleeding that required unplanned medical or surgical treatment or unplanned laboratory evaluation even if it did not meet the criteria for TIMI major or minor bleeding. The Kaplan-Meier estimate reports the percentage of participants who experienced clinically significant bleeding within 3 years from randomization.
Time Frame: up to 3 years
Population: as for outcome 19
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 10049 | 10059
Percentage of Participants | 11.1 | 15.2
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p < 0.001, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 1.42, 95% CI 2-sided [1.31 to 1.54] — [estimate comment as in outcome 1, analysis 1]

21. Post Hoc Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced Death From Any Cause, MI, Stroke, or UCR Within 3 Years From Randomization
Description: as for outcome 5
Time Frame: up to 3 years
Population: Intended Label Population: all enrolled participants with CAD or PAD and no history of a stroke or TIA
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 10090 | 10080
Percentage of Participants | 13.5 | 11.9
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p < 0.001, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.86, 95% CI 2-sided [0.79 to 0.93] — [estimate comment as in outcome 1, analysis 1]

22. Post Hoc Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced CV Death or an MI Within 3 Years From Randomization
Description: The time (in days) from study start to the occurrence of CV death or first occurrence of an MI. A CEC reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). If a participant had a fatal event that was not part of a specific endpoint for analysis, they were censored at the time of death. The Kaplan-Meier estimate reports the percentage of participants who experienced CV death or MI within 3 years from randomization.
Time Frame: up to 3 years
Population: Intended Label Population: all enrolled participants with CAD or PAD and no history of a stroke or TIA
Measure: Number; unit: Percentage of Partcipants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 10090 | 10080
Percentage of Partcipants | 8.3 | 7.2
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p < 0.001, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.83, 95% CI 2-sided [0.75 to 0.93] — [estimate comment as in outcome 1, analysis 1]

23. Post Hoc Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced CV Death, MI, Stroke, UCR, or UH-VCIN Within 3 Years From Randomization
Description: The time (in days) from study start to the first occurrence of any of the following clinical outcomes was recorded: CV death, MI, stroke, UCR, or UH-VCIN . A CEC reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). If a participant had a fatal event that was not part of a specific endpoint for analysis, they were censored at the time of death. The Kaplan-Meier estimate reports the percentage of participants who experienced CV death, MI, stroke, UCR, or UH-VCIN within 3 years from randomization.
Time Frame: up to 3 years
Population: Intended Label Population: all enrolled participants with CAD or PAD and no history of a stroke or TIA
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 10090 | 10080
Percentage of Participants | 13.9 | 11.9
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p < 0.001, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.83, 95% CI 2-sided [0.77 to 0.90] — [estimate comment as in outcome 1, analysis 1]

24. Post Hoc Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Died From Any Cause, or Experienced an MI, Stroke, or Any Revascularization Within 3 Years From Randomization
Description: as for outcome 8
Time Frame: up to 3 years
Population: Intended Label Population: all enrolled participants with CAD or PAD and no history of a stroke or TIA
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 10090 | 10080
Percentage of Participants | 22.5 | 20.1
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p < 0.001, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.89, 95% CI 2-sided [0.83 to 0.95] — [estimate comment as in outcome 1, analysis 1]

25. Post Hoc Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced CV Death, MI, Stroke, Any Revascularization, or UH-VCIN Within 3 Years From Randomization
Description: as for outcome 9
Time Frame: up to 3 years
Population: Intended Label Population: all enrolled participants with CAD or PAD and no history of a stroke or TIA
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 10090 | 10080
Percentage of Participants | 21.8 | 19.3
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p < 0.001, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.88, 95% CI 2-sided [0.83 to 0.94] — [estimate comment as in outcome 1, analysis 1]

26. Post Hoc Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced CV Death Within 3 Years From Randomization
Description: The time (in days) from study start to the CV death (if reported) was recorded. A CEC reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). If a participant had a fatal event that was not part of a specific endpoint for analysis, they were censored at the time of death. The Kaplan-Meier estimate reports the percentage of participants who experienced CV death within 3 years from randomization.
Time Frame: up to 3 years
Population: Intended Label Population: all enrolled participants with CAD or PAD and no history of a stroke or TIA
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 10090 | 10080
Percentage of Participants | 2.8 | 2.4
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p = 0.108, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.86, 95% CI 2-sided [0.71 to 1.03] — [estimate comment as in outcome 1, analysis 1]

27. Post Hoc Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced an MI Within 3 Years From Randomization
Description: as for outcome 11
Time Frame: up to 3 years
Population: Intended Label Population: all enrolled participants with CAD or PAD and no history of a stroke or TIA
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 10090 | 10080
Percentage of Participants | 6.4 | 5.4
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p = 0.002, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.82, 95% CI 2-sided [0.73 to 0.93] — [estimate comment as in outcome 1, analysis 1]

28. Post Hoc Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced UCR Within 3 Years From Randomization
Description: as for outcome 12
Time Frame: up to 3 years
Population: Intended Label Population: all enrolled participants with CAD or PAD and no history of a stroke or TIA
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 10090 | 10080
Percentage of Participants | 3.0 | 2.8
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p = 0.127, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.88, 95% CI 2-sided [0.74 to 1.04] — [estimate comment as in outcome 1, analysis 1]

29. Post Hoc Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Experienced a Stroke Within 3 Years From Randomization
Description: as for outcome 13
Time Frame: up to 3 years
Population: Intended Label Population: all enrolled participants with CAD or PAD and no history of a stroke or TIA
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 10090 | 10080
Percentage of Participants | 1.6 | 1.2
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p = 0.002, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.67, 95% CI 2-sided [0.52 to 0.87] — [estimate comment as in outcome 1, analysis 1]

30. Post Hoc Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Died From Any Cause Within 3 Years From Randomization
Description: as for outcome 14
Time Frame: up to 3 years
Population: Intended Label Population: all enrolled participants with CAD or PAD and no history of a stroke or TIA
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 10090 | 10080
Percentage of Participants | 4.8 | 4.5
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p = 0.249, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.92, 95% CI 2-sided [0.80 to 1.06] — [estimate comment as in outcome 1, analysis 1]

31. Post Hoc Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Had a UH-VCIN Within 3 Years From Randomization
Description: The time (in days) from study start to the first occurrence of a UH-VCIN was recorded. A CEC reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). If a participant had a fatal event that was not part of a specific endpoint for analysis, they were censored at the time of death. The Kaplan-Meier estimate reports the percentage of participants who had a UH-VCIN within 3 years from randomization.
Time Frame: up to 3 years
Population: Intended Label Population: all enrolled participants with CAD or PAD and no history of a stroke or TIA
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 10090 | 10080
Percentage of Participants | 5.6 | 4.9
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p = 0.019, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.86, 95% CI 2-sided [0.76 to 0.98] — [estimate comment as in outcome 1, analysis 1]

32. Post Hoc Outcome: Kaplan-Meier Estimate of the Percentage of Participants Who Had Any Revascularization Performed Within 3 Years From Randomization
Description: The time (in days) from study start to the first occurrence of any revascularization was recorded. A CEC reviewed and adjudicated each suspected efficacy endpoint event while blinded to treatment. Participants who did not have any endpoint event until last visit or participants who were lost to follow-up and had no event were censored at the time of last available information (last study visit). If a participant had a fatal event that was not part of a specific endpoint for analysis, they were censored at the time of death. The Kaplan-Meier estimate reports the percentage of participants who had any revascularization performed within 3 years from randomization.
Time Frame: up to 3 years
Population: Intended Label Population: all enrolled participants with CAD or PAD and no history of a stroke or TIA
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Vorapaxar
Number analyzed (Participants) | 10090 | 10080
Percentage of Participants | 16.6 | 14.7
Statistical Analysis 1: Comparison: Placebo vs Vorapaxar; Test type: Superiority or Other; p = 0.003, Cox Proportional Hazards Regression; Hazard Ratio calculated with covariates for treatment and stratification factors; Cox Proportional Hazard = 0.89, 95% CI 2-sided [0.83 to 0.96] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: up to 3 years
Description: Adverse events are reported using the As Treated Population, which included all participants who received at least 1 dose of study medication and are reported according to treatment received
Arm/Group | Placebo | Vorapaxar
Serious Adverse Events (participants affected / at risk) | 3419/13166 | 3514/13186
Other Adverse Events (participants affected / at risk) | 2280/13166 | 2541/13186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=13166) | Vorapaxar (N=13186)
ANAEMIA (Blood and lymphatic system disorders) | 12 (13) | 45 (47)
ANAEMIA HAEMOLYTIC AUTOIMMUNE (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
ANAEMIA OF CHRONIC DISEASE (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
APLASIA PURE RED CELL (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
AUTOIMMUNE THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
COAGULOPATHY (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
HAEMORRHAGIC DIATHESIS (Blood and lymphatic system disorders) | 4 (4) | 7 (7)
HEPARIN-INDUCED THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
IDIOPATHIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 4 (4) | 16 (16)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
MICROCYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
NEPHROGENIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
NORMOCHROMIC NORMOCYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
PANCYTOPENIA (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
PERNICIOUS ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
RETROPERITONEAL LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
SPLENIC HAEMORRHAGE (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 23 (23) | 19 (20)
THROMBOCYTOSIS (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
THROMBOTIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 (0) | 1 (1)
ADAMS-STOKES SYNDROME (Cardiac disorders) | 0 (0) | 1 (1)
ANGINA PECTORIS (Cardiac disorders) | 7 (8) | 2 (2)
AORTIC VALVE INCOMPETENCE (Cardiac disorders) | 1 (1) | 1 (1)
AORTIC VALVE STENOSIS (Cardiac disorders) | 4 (4) | 5 (5)
ARRHYTHMIA (Cardiac disorders) | 2 (2) | 3 (3)
ARRHYTHMIA SUPRAVENTRICULAR (Cardiac disorders) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 106 (118) | 137 (156)
ATRIAL FLUTTER (Cardiac disorders) | 18 (19) | 28 (28)
ATRIAL TACHYCARDIA (Cardiac disorders) | 3 (3) | 0 (0)
ATRIAL THROMBOSIS (Cardiac disorders) | 1 (1) | 2 (2)
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 3 (3) | 3 (3)
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 13 (13) | 19 (19)
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 0 (0) | 1 (1)
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 8 (9) | 4 (4)
BIFASCICULAR BLOCK (Cardiac disorders) | 1 (1) | 0 (0)
BRADYCARDIA (Cardiac disorders) | 27 (27) | 20 (20)
BUNDLE BRANCH BLOCK LEFT (Cardiac disorders) | 2 (3) | 0 (0)
BUNDLE BRANCH BLOCK RIGHT (Cardiac disorders) | 2 (2) | 0 (0)
CARDIAC ANEURYSM (Cardiac disorders) | 0 (0) | 2 (2)
CARDIAC ARREST (Cardiac disorders) | 13 (13) | 2 (2)
CARDIAC ASTHMA (Cardiac disorders) | 0 (0) | 2 (2)
CARDIAC FAILURE (Cardiac disorders) | 174 (222) | 183 (245)
CARDIAC FAILURE ACUTE (Cardiac disorders) | 5 (5) | 4 (5)
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 1 (1) | 1 (1)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 82 (99) | 95 (121)
CARDIAC TAMPONADE (Cardiac disorders) | 5 (5) | 4 (5)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 4 (4) | 3 (3)
CARDIOGENIC SHOCK (Cardiac disorders) | 10 (10) | 8 (8)
CARDIOMYOPATHY (Cardiac disorders) | 5 (5) | 3 (3)
CARDIOPULMONARY FAILURE (Cardiac disorders) | 1 (1) | 0 (0)
CHRONOTROPIC INCOMPETENCE (Cardiac disorders) | 1 (1) | 0 (0)
CONDUCTION DISORDER (Cardiac disorders) | 2 (2) | 0 (0)
CONGESTIVE CARDIOMYOPATHY (Cardiac disorders) | 1 (1) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (1) | 1 (1)
DRESSLER'S SYNDROME (Cardiac disorders) | 1 (1) | 2 (3)
EXTRASYSTOLES (Cardiac disorders) | 2 (2) | 0 (0)
HEART VALVE INCOMPETENCE (Cardiac disorders) | 1 (1) | 0 (0)
HYPERTENSIVE HEART DISEASE (Cardiac disorders) | 1 (1) | 0 (0)
INTRACARDIAC THROMBUS (Cardiac disorders) | 3 (3) | 1 (1)
ISCHAEMIC CARDIOMYOPATHY (Cardiac disorders) | 8 (8) | 11 (11)
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 2 (2) | 10 (10)
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 0 (0) | 2 (2)
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 4 (4) | 4 (4)
MITRAL VALVE PROLAPSE (Cardiac disorders) | 1 (1) | 0 (0)
MITRAL VALVE STENOSIS (Cardiac disorders) | 1 (1) | 3 (3)
MYOCARDIAL RUPTURE (Cardiac disorders) | 2 (2) | 0 (0)
MYOPERICARDITIS (Cardiac disorders) | 0 (0) | 1 (1)
NODAL ARRHYTHMIA (Cardiac disorders) | 1 (1) | 2 (2)
PALPITATIONS (Cardiac disorders) | 3 (3) | 7 (7)
PERICARDIAL EFFUSION (Cardiac disorders) | 4 (4) | 3 (3)
PERICARDIAL HAEMORRHAGE (Cardiac disorders) | 2 (2) | 8 (8)
PERICARDITIS (Cardiac disorders) | 9 (9) | 3 (3)
PULSELESS ELECTRICAL ACTIVITY (Cardiac disorders) | 1 (1) | 3 (3)
SICK SINUS SYNDROME (Cardiac disorders) | 20 (20) | 20 (22)
SINUS ARREST (Cardiac disorders) | 1 (1) | 1 (1)
SINUS ARRHYTHMIA (Cardiac disorders) | 4 (4) | 4 (4)
SINUS BRADYCARDIA (Cardiac disorders) | 4 (4) | 3 (3)
SINUS TACHYCARDIA (Cardiac disorders) | 4 (4) | 4 (4)
STRESS CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 1 (2)
SUPRAVENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1 (1) | 1 (1)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 16 (20) | 13 (14)
TACHYARRHYTHMIA (Cardiac disorders) | 2 (2) | 1 (1)
TACHYCARDIA (Cardiac disorders) | 1 (1) | 2 (2)
TORSADE DE POINTES (Cardiac disorders) | 0 (0) | 2 (2)
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 2 (2) | 3 (3)
VENTRICULAR ASYSTOLE (Cardiac disorders) | 0 (0) | 1 (1)
VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 (0) | 1 (1)
VENTRICULAR DYSSYNCHRONY (Cardiac disorders) | 1 (1) | 0 (0)
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 4 (5) | 4 (4)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 15 (16) | 16 (16)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 37 (49) | 37 (42)
ARTERIOVENOUS MALFORMATION (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
ATRIAL SEPTAL DEFECT (Congenital, familial and genetic disorders) | 0 (0) | 2 (2)
EPIDERMOLYSIS (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL ANGIODYSPLASIA (Congenital, familial and genetic disorders) | 0 (0) | 2 (2)
GASTROINTESTINAL ANGIODYSPLASIA HAEMORRHAGIC (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL ARTERIOVENOUS MALFORMATION (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
HAEMORRHAGIC ARTERIOVENOUS MALFORMATION (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
HIP DYSPLASIA (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
HYDROCELE (Congenital, familial and genetic disorders) | 2 (2) | 0 (0)
PHIMOSIS (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
PORPHYRIA (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
PYLORIC STENOSIS (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
VENTRICULAR SEPTAL DEFECT (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
ACUTE VESTIBULAR SYNDROME (Ear and labyrinth disorders) | 1 (1) | 0 (0)
DEAFNESS (Ear and labyrinth disorders) | 1 (1) | 0 (0)
HYPOACUSIS (Ear and labyrinth disorders) | 0 (0) | 2 (2)
MENIERE'S DISEASE (Ear and labyrinth disorders) | 3 (3) | 0 (0)
SUDDEN HEARING LOSS (Ear and labyrinth disorders) | 2 (2) | 1 (1)
VERTIGO (Ear and labyrinth disorders) | 16 (17) | 23 (24)
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 5 (5) | 3 (3)
VESTIBULAR DISORDER (Ear and labyrinth disorders) | 0 (0) | 2 (2)
ADDISON'S DISEASE (Endocrine disorders) | 0 (0) | 1 (1)
ADRENAL MASS (Endocrine disorders) | 0 (0) | 1 (1)
AUTOIMMUNE THYROIDITIS (Endocrine disorders) | 1 (1) | 1 (1)
BASEDOW'S DISEASE (Endocrine disorders) | 1 (1) | 1 (1)
GOITRE (Endocrine disorders) | 5 (5) | 1 (1)
HYPERCALCAEMIA OF MALIGNANCY (Endocrine disorders) | 1 (1) | 0 (0)
HYPERPARATHYROIDISM (Endocrine disorders) | 1 (1) | 0 (0)
HYPERTHYROIDISM (Endocrine disorders) | 3 (3) | 4 (4)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 1 (1)
INAPPROPRIATE ANTIDIURETIC HORMONE SECRETION (Endocrine disorders) | 2 (2) | 0 (0)
AMAUROSIS (Eye disorders) | 0 (0) | 1 (1)
BLINDNESS UNILATERAL (Eye disorders) | 1 (1) | 0 (0)
CATARACT (Eye disorders) | 15 (15) | 10 (12)
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 0 (0) | 2 (2)
CORNEAL OEDEMA (Eye disorders) | 1 (1) | 0 (0)
DIABETIC RETINOPATHY (Eye disorders) | 2 (2) | 2 (3)
ENDOCRINE OPHTHALMOPATHY (Eye disorders) | 0 (0) | 1 (1)
EYE HAEMORRHAGE (Eye disorders) | 5 (6) | 3 (3)
GLAUCOMA (Eye disorders) | 3 (3) | 1 (1)
HYPHAEMA (Eye disorders) | 0 (0) | 1 (1)
LACRIMATION INCREASED (Eye disorders) | 0 (0) | 1 (1)
MACULAR DEGENERATION (Eye disorders) | 0 (0) | 1 (1)
MACULAR FIBROSIS (Eye disorders) | 1 (1) | 0 (0)
MACULAR HOLE (Eye disorders) | 0 (0) | 1 (1)
OCULAR HYPERTENSION (Eye disorders) | 0 (0) | 1 (1)
OPTIC ISCHAEMIC NEUROPATHY (Eye disorders) | 1 (1) | 0 (0)
OPTIC NEUROPATHY (Eye disorders) | 1 (1) | 0 (0)
POSTERIOR CAPSULE OPACIFICATION (Eye disorders) | 1 (1) | 0 (0)
RETINAL ARTERY THROMBOSIS (Eye disorders) | 0 (0) | 1 (1)
RETINAL DETACHMENT (Eye disorders) | 6 (6) | 4 (4)
RETINAL VEIN OCCLUSION (Eye disorders) | 0 (0) | 1 (1)
RETINAL VEIN THROMBOSIS (Eye disorders) | 0 (0) | 1 (1)
ULCERATIVE KERATITIS (Eye disorders) | 1 (1) | 0 (0)
VISION BLURRED (Eye disorders) | 0 (0) | 1 (1)
VISUAL IMPAIRMENT (Eye disorders) | 0 (0) | 1 (1)
VITREOUS HAEMORRHAGE (Eye disorders) | 2 (2) | 0 (0)
ABDOMINAL ADHESIONS (Gastrointestinal disorders) | 1 (1) | 2 (2)
ABDOMINAL COMPARTMENT SYNDROME (Gastrointestinal disorders) | 1 (1) | 0 (0)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 (1) | 1 (1)
ABDOMINAL HERNIA (Gastrointestinal disorders) | 6 (6) | 4 (4)
ABDOMINAL HERNIA OBSTRUCTIVE (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL MASS (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 17 (18) | 9 (9)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 9 (9) | 10 (10)
ABDOMINAL WALL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
ACUTE ABDOMEN (Gastrointestinal disorders) | 2 (2) | 0 (0)
ANAL FISTULA (Gastrointestinal disorders) | 2 (2) | 2 (2)
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (2) | 2 (2)
ASCITES (Gastrointestinal disorders) | 2 (2) | 1 (1)
BARRETT'S OESOPHAGUS (Gastrointestinal disorders) | 2 (2) | 1 (1)
BUCCAL POLYP (Gastrointestinal disorders) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 7 (7) | 9 (9)
COLITIS EROSIVE (Gastrointestinal disorders) | 0 (0) | 1 (1)
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 8 (8) | 8 (9)
COLITIS ULCERATIVE (Gastrointestinal disorders) | 1 (1) | 2 (2)
COLONIC POLYP (Gastrointestinal disorders) | 6 (6) | 14 (14)
COLONIC PSEUDO-OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 10 (10) | 11 (11)
CROHN'S DISEASE (Gastrointestinal disorders) | 3 (3) | 3 (3)
DENTAL CARIES (Gastrointestinal disorders) | 1 (1) | 1 (1)
DENTAL NECROSIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
DIABETIC GASTROPARESIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 4 (4) | 7 (8)
DIARRHOEA HAEMORRHAGIC (Gastrointestinal disorders) | 2 (2) | 2 (2)
DIVERTICULAR PERFORATION (Gastrointestinal disorders) | 2 (2) | 0 (0)
DIVERTICULITIS INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 1 (1) | 1 (1)
DIVERTICULUM (Gastrointestinal disorders) | 3 (3) | 4 (4)
DIVERTICULUM INTESTINAL (Gastrointestinal disorders) | 0 (0) | 2 (2)
DIVERTICULUM INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 0 (0) | 3 (5)
DIVERTICULUM OESOPHAGEAL (Gastrointestinal disorders) | 1 (1) | 1 (1)
DUODENAL PERFORATION (Gastrointestinal disorders) | 2 (2) | 0 (0)
DUODENAL ULCER (Gastrointestinal disorders) | 5 (5) | 8 (9)
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 3 (3) | 3 (3)
DUODENITIS (Gastrointestinal disorders) | 2 (2) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 5 (5) | 10 (10)
DYSPHAGIA (Gastrointestinal disorders) | 5 (5) | 4 (4)
ENTERITIS (Gastrointestinal disorders) | 4 (4) | 2 (2)
ENTEROCELE (Gastrointestinal disorders) | 1 (1) | 0 (0)
ENTEROCOLITIS (Gastrointestinal disorders) | 1 (1) | 1 (1)
ENTEROCOLITIS HAEMORRHAGIC (Gastrointestinal disorders) | 1 (1) | 0 (0)
ENTEROVESICAL FISTULA (Gastrointestinal disorders) | 1 (1) | 0 (0)
EPIGASTRIC DISCOMFORT (Gastrointestinal disorders) | 1 (1) | 0 (0)
EPIPLOIC APPENDAGITIS (Gastrointestinal disorders) | 1 (1) | 1 (1)
EROSIVE DUODENITIS (Gastrointestinal disorders) | 1 (1) | 1 (1)
EROSIVE OESOPHAGITIS (Gastrointestinal disorders) | 3 (3) | 4 (4)
FAECALOMA (Gastrointestinal disorders) | 4 (4) | 2 (2)
FAECES DISCOLOURED (Gastrointestinal disorders) | 1 (1) | 0 (0)
FEMORAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 1 (1) | 0 (0)
FOOD POISONING (Gastrointestinal disorders) | 1 (1) | 1 (1)
FUNCTIONAL GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC DISORDER (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 1 (2) | 3 (3)
GASTRIC PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRIC ULCER (Gastrointestinal disorders) | 6 (6) | 11 (11)
GASTRIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 5 (5) | 6 (6)
GASTRIC ULCER PERFORATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRIC VOLVULUS (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 29 (29) | 26 (26)
GASTRITIS ALCOHOLIC (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTRITIS ATROPHIC (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTRITIS EROSIVE (Gastrointestinal disorders) | 3 (3) | 6 (7)
GASTRODUODENAL ULCER (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 0 (0) | 1 (1)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 38 (42) | 62 (70)
GASTROINTESTINAL INFLAMMATION (Gastrointestinal disorders) | 2 (2) | 0 (0)
GASTROINTESTINAL NECROSIS (Gastrointestinal disorders) | 0 (0) | 3 (3)
GASTROINTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 (2) | 1 (1)
GASTROINTESTINAL TELANGIECTASIA (Gastrointestinal disorders) | 0 (0) | 2 (2)
GASTROINTESTINAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 2 (2) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 31 (33) | 23 (24)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 (0) | 2 (2)
HAEMATEMESIS (Gastrointestinal disorders) | 19 (19) | 28 (28)
HAEMATOCHEZIA (Gastrointestinal disorders) | 21 (24) | 16 (18)
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 5 (6) | 7 (7)
HAEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 4 (4)
HERNIAL EVENTRATION (Gastrointestinal disorders) | 1 (2) | 0 (0)
HIATUS HERNIA (Gastrointestinal disorders) | 5 (5) | 4 (4)
ILEAL STENOSIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
ILEUS (Gastrointestinal disorders) | 5 (5) | 8 (10)
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 2 (2) | 2 (2)
INFLAMMATORY BOWEL DISEASE (Gastrointestinal disorders) | 0 (0) | 1 (1)
INGUINAL HERNIA (Gastrointestinal disorders) | 35 (35) | 42 (44)
INGUINAL HERNIA STRANGULATED (Gastrointestinal disorders) | 1 (1) | 0 (0)
INGUINAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 2 (2) | 4 (4)
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 8 (8) | 3 (3)
INTESTINAL MASS (Gastrointestinal disorders) | 0 (0) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 9 (9) | 13 (14)
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 (1) | 7 (7)
INTESTINAL POLYP (Gastrointestinal disorders) | 1 (1) | 2 (2)
INTESTINAL STRANGULATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
JEJUNAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
LARGE INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 1 (1)
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
LARGE INTESTINAL ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
LARGE INTESTINAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 2 (2) | 4 (4)
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 8 (8) | 5 (5)
LUMBAR HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
MALABSORPTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
MALLORY-WEISS SYNDROME (Gastrointestinal disorders) | 2 (2) | 2 (2)
MECHANICAL ILEUS (Gastrointestinal disorders) | 1 (1) | 1 (1)
MELAENA (Gastrointestinal disorders) | 44 (49) | 69 (76)
MESENTERIC ARTERY STENOSIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
MESENTERIC ARTERY THROMBOSIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
MESENTERIC VASCULAR INSUFFICIENCY (Gastrointestinal disorders) | 0 (0) | 1 (1)
MOUTH CYST (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 5 (5) | 8 (8)
OESOPHAGEAL ACHALASIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
OESOPHAGEAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
OESOPHAGEAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0)
OESOPHAGEAL RUPTURE (Gastrointestinal disorders) | 0 (0) | 2 (2)
OESOPHAGEAL SPASM (Gastrointestinal disorders) | 1 (1) | 1 (1)
OESOPHAGEAL STENOSIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
OESOPHAGEAL ULCER (Gastrointestinal disorders) | 0 (0) | 2 (2)
OESOPHAGEAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
OESOPHAGITIS (Gastrointestinal disorders) | 4 (4) | 10 (11)
PANCREATIC CYST (Gastrointestinal disorders) | 1 (1) | 0 (0)
PANCREATIC DISORDER (Gastrointestinal disorders) | 1 (1) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 17 (21) | 17 (18)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 11 (13) | 9 (11)
PANCREATITIS RELAPSING (Gastrointestinal disorders) | 1 (1) | 0 (0)
PAPILLA OF VATER STENOSIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
PAROTID GLAND ENLARGEMENT (Gastrointestinal disorders) | 1 (1) | 0 (0)
PEPTIC ULCER (Gastrointestinal disorders) | 2 (2) | 5 (5)
PEPTIC ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 2 (2)
PERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 2 (2)
PHARYNGOESOPHAGEAL DIVERTICULUM (Gastrointestinal disorders) | 1 (1) | 0 (0)
POLYP COLORECTAL (Gastrointestinal disorders) | 0 (0) | 1 (1)
PROCTITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
PROCTITIS HAEMORRHAGIC (Gastrointestinal disorders) | 1 (1) | 0 (0)
PROCTITIS ULCERATIVE (Gastrointestinal disorders) | 1 (1) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 37 (41) | 53 (59)
RECTAL PROLAPSE (Gastrointestinal disorders) | 0 (0) | 1 (1)
RECTAL ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0)
RETROPERITONEAL HAEMATOMA (Gastrointestinal disorders) | 0 (0) | 2 (2)
RETROPERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 3 (3) | 8 (8)
SALIVARY GLAND CALCULUS (Gastrointestinal disorders) | 1 (1) | 0 (0)
SMALL INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 (2) | 2 (2)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 14 (18) | 12 (12)
SMALL INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 (1) | 1 (1)
SPIGELIAN HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
SPLENIC ARTERY ANEURYSM (Gastrointestinal disorders) | 1 (1) | 0 (0)
SUBILEUS (Gastrointestinal disorders) | 1 (1) | 1 (1)
THROMBOSIS MESENTERIC VESSEL (Gastrointestinal disorders) | 1 (1) | 0 (0)
TONGUE HAEMATOMA (Gastrointestinal disorders) | 1 (1) | 0 (0)
TONGUE OEDEMA (Gastrointestinal disorders) | 1 (1) | 0 (0)
UMBILICAL HERNIA (Gastrointestinal disorders) | 10 (10) | 6 (6)
UMBILICAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 2 (2) | 2 (2)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 17 (20) | 15 (16)
VARICES OESOPHAGEAL (Gastrointestinal disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 4 (4) | 1 (1)
ADVERSE DRUG REACTION (General disorders) | 12 (12) | 16 (16)
APPLICATION SITE BLEEDING (General disorders) | 1 (1) | 0 (0)
ASTHENIA (General disorders) | 5 (5) | 1 (1)
CATHETER SITE HAEMATOMA (General disorders) | 4 (4) | 8 (8)
CATHETER SITE HAEMORRHAGE (General disorders) | 5 (5) | 5 (5)
CHEST DISCOMFORT (General disorders) | 10 (11) | 6 (6)
CHEST PAIN (General disorders) | 14 (16) | 15 (15)
CYST (General disorders) | 0 (0) | 1 (1)
CYST RUPTURE (General disorders) | 1 (1) | 0 (0)
DEVICE BREAKAGE (General disorders) | 0 (0) | 1 (1)
DEVICE DISLOCATION (General disorders) | 2 (3) | 3 (4)
DEVICE FAILURE (General disorders) | 0 (0) | 2 (2)
DEVICE LEAD DAMAGE (General disorders) | 1 (1) | 2 (2)
DEVICE MALFUNCTION (General disorders) | 3 (3) | 7 (7)
DEVICE OCCLUSION (General disorders) | 1 (1) | 1 (1)
DISCOMFORT (General disorders) | 2 (2) | 0 (0)
DRUG INTERACTION (General disorders) | 0 (0) | 1 (1)
EXERCISE TOLERANCE DECREASED (General disorders) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 2 (2)
GAIT DISTURBANCE (General disorders) | 2 (2) | 2 (2)
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 (1) | 1 (1)
GRAVITATIONAL OEDEMA (General disorders) | 1 (1) | 0 (0)
HERNIA (General disorders) | 2 (2) | 2 (3)
HERNIA OBSTRUCTIVE (General disorders) | 0 (0) | 2 (2)
HYPERPLASIA (General disorders) | 0 (0) | 1 (1)
HYPERTROPHY (General disorders) | 1 (1) | 0 (0)
HYPOTHERMIA (General disorders) | 1 (1) | 0 (0)
ILL-DEFINED DISORDER (General disorders) | 1 (1) | 0 (0)
IMPAIRED HEALING (General disorders) | 5 (5) | 6 (6)
IMPLANT SITE EROSION (General disorders) | 1 (1) | 0 (0)
IMPLANT SITE PAIN (General disorders) | 0 (0) | 1 (1)
INFLAMMATION (General disorders) | 2 (2) | 0 (0)
MALAISE (General disorders) | 4 (4) | 0 (0)
MEDICAL DEVICE COMPLICATION (General disorders) | 1 (1) | 1 (1)
MUCOSAL INFLAMMATION (General disorders) | 1 (1) | 0 (0)
MULTI-ORGAN DISORDER (General disorders) | 0 (0) | 2 (2)
MULTI-ORGAN FAILURE (General disorders) | 4 (4) | 6 (6)
NECROSIS (General disorders) | 1 (1) | 0 (0)
NODULE (General disorders) | 1 (1) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 458 (548) | 443 (519)
OEDEMA (General disorders) | 0 (0) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 4 (4) | 4 (4)
PAIN (General disorders) | 1 (1) | 1 (1)
PERFORATED ULCER (General disorders) | 1 (2) | 0 (0)
POLYP (General disorders) | 1 (1) | 3 (3)
POLYSEROSITIS (General disorders) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 11 (12) | 9 (9)
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 2 (2) | 0 (0)
THROMBOSIS IN DEVICE (General disorders) | 1 (1) | 0 (0)
ULCER (General disorders) | 0 (0) | 1 (1)
ULCER HAEMORRHAGE (General disorders) | 2 (2) | 1 (1)
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 0 (0) | 1 (1)
BILE DUCT STONE (Hepatobiliary disorders) | 6 (6) | 4 (4)
BILIARY COLIC (Hepatobiliary disorders) | 2 (2) | 3 (3)
BILIARY DILATATION (Hepatobiliary disorders) | 0 (0) | 1 (1)
BILIARY DYSKINESIA (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLANGITIS (Hepatobiliary disorders) | 1 (1) | 3 (3)
CHOLANGITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 26 (26) | 31 (32)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 18 (19) | 18 (18)
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 1 (1) | 3 (3)
CHOLELITHIASIS (Hepatobiliary disorders) | 42 (42) | 42 (43)
CHOLESTASIS (Hepatobiliary disorders) | 2 (2) | 0 (0)
GALLBLADDER DISORDER (Hepatobiliary disorders) | 1 (1) | 0 (0)
GALLBLADDER POLYP (Hepatobiliary disorders) | 1 (1) | 1 (1)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 5 (5) | 1 (1)
HEPATIC FAILURE (Hepatobiliary disorders) | 1 (1) | 3 (3)
HEPATIC MASS (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATIC STEATOSIS (Hepatobiliary disorders) | 1 (1) | 1 (1)
HEPATITIS (Hepatobiliary disorders) | 1 (1) | 1 (1)
HEPATITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 1 (1)
HEPATITIS TOXIC (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATORENAL SYNDROME (Hepatobiliary disorders) | 0 (0) | 1 (1)
HEPATOTOXICITY (Hepatobiliary disorders) | 1 (1) | 0 (0)
ISCHAEMIC HEPATITIS (Hepatobiliary disorders) | 1 (1) | 1 (1)
LIVER DISORDER (Hepatobiliary disorders) | 1 (1) | 0 (0)
ALLERGY TO ARTHROPOD STING (Immune system disorders) | 1 (1) | 1 (1)
ANAPHYLACTIC REACTION (Immune system disorders) | 1 (1) | 2 (2)
ANAPHYLACTIC SHOCK (Immune system disorders) | 2 (2) | 1 (1)
DRUG HYPERSENSITIVITY (Immune system disorders) | 10 (10) | 4 (4)
FOOD ALLERGY (Immune system disorders) | 1 (1) | 0 (0)
HYPERSENSITIVITY (Immune system disorders) | 6 (6) | 1 (1)
HYPOGAMMAGLOBULINAEMIA (Immune system disorders) | 1 (1) | 0 (0)
ABDOMINAL ABSCESS (Infections and infestations) | 1 (1) | 2 (2)
ABDOMINAL WALL ABSCESS (Infections and infestations) | 0 (0) | 2 (2)
ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
ABSCESS INTESTINAL (Infections and infestations) | 1 (1) | 0 (0)
ABSCESS LIMB (Infections and infestations) | 4 (4) | 7 (7)
ABSCESS ORAL (Infections and infestations) | 0 (0) | 1 (1)
ANAL ABSCESS (Infections and infestations) | 3 (4) | 6 (7)
APPENDICEAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
APPENDICITIS (Infections and infestations) | 23 (23) | 20 (20)
ARTERIOVENOUS FISTULA SITE INFECTION (Infections and infestations) | 0 (0) | 1 (1)
ARTERIOVENOUS GRAFT SITE ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
ARTERIOVENOUS GRAFT SITE INFECTION (Infections and infestations) | 1 (1) | 1 (1)
ARTHRITIS BACTERIAL (Infections and infestations) | 2 (2) | 2 (2)
ARTHRITIS INFECTIVE (Infections and infestations) | 2 (2) | 0 (0)
ASPERGILLOMA (Infections and infestations) | 1 (1) | 0 (0)
BACTERAEMIA (Infections and infestations) | 2 (2) | 3 (3)
BACTERIAL INFECTION (Infections and infestations) | 0 (0) | 3 (3)
BACTERIAL PROSTATITIS (Infections and infestations) | 0 (0) | 1 (1)
BILIARY SEPSIS (Infections and infestations) | 0 (0) | 1 (1)
BLASTOCYSTIS INFECTION (Infections and infestations) | 1 (1) | 0 (0)
BORRELIA INFECTION (Infections and infestations) | 0 (0) | 1 (1)
BRONCHIOLITIS (Infections and infestations) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 29 (29) | 27 (27)
BRONCHITIS BACTERIAL (Infections and infestations) | 2 (2) | 1 (1)
BRONCHOPNEUMONIA (Infections and infestations) | 10 (10) | 12 (12)
BURSITIS INFECTIVE (Infections and infestations) | 1 (1) | 2 (2)
CAMPYLOBACTER GASTROENTERITIS (Infections and infestations) | 1 (1) | 2 (2)
CAMPYLOBACTER INTESTINAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
CARDIAC INFECTION (Infections and infestations) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 38 (41) | 42 (45)
CELLULITIS OF MALE EXTERNAL GENITAL ORGAN (Infections and infestations) | 0 (0) | 1 (1)
CENTRAL NERVOUS SYSTEM INFECTION (Infections and infestations) | 1 (1) | 1 (1)
CHOLECYSTITIS INFECTIVE (Infections and infestations) | 2 (2) | 2 (2)
CHRONIC SINUSITIS (Infections and infestations) | 1 (1) | 2 (2)
CLOSTRIDIAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
CLOSTRIDIUM COLITIS (Infections and infestations) | 0 (0) | 1 (1)
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 16 (18) | 4 (4)
COCCIDIOIDOMYCOSIS (Infections and infestations) | 0 (0) | 1 (1)
CYSTITIS (Infections and infestations) | 2 (2) | 7 (7)
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 1 (1) | 0 (0)
DENGUE FEVER (Infections and infestations) | 0 (0) | 2 (2)
DEVICE RELATED INFECTION (Infections and infestations) | 7 (9) | 5 (5)
DEVICE RELATED SEPSIS (Infections and infestations) | 1 (2) | 0 (0)
DIABETIC FOOT INFECTION (Infections and infestations) | 4 (5) | 3 (3)
DIABETIC GANGRENE (Infections and infestations) | 0 (0) | 1 (1)
DISSEMINATED TUBERCULOSIS (Infections and infestations) | 0 (0) | 1 (1)
DIVERTICULITIS (Infections and infestations) | 20 (21) | 16 (17)
DYSENTERY (Infections and infestations) | 0 (0) | 1 (1)
EAR INFECTION (Infections and infestations) | 1 (1) | 0 (0)
ECZEMA INFECTED (Infections and infestations) | 1 (1) | 0 (0)
EMPYEMA (Infections and infestations) | 1 (1) | 1 (1)
ENCEPHALITIS HERPES (Infections and infestations) | 0 (0) | 1 (1)
ENDOCARDITIS (Infections and infestations) | 1 (1) | 2 (2)
ENDOPHTHALMITIS (Infections and infestations) | 0 (0) | 1 (1)
ENTERITIS INFECTIOUS (Infections and infestations) | 0 (0) | 1 (1)
ENTEROBACTER INFECTION (Infections and infestations) | 0 (0) | 1 (1)
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 1 (1) | 0 (0)
EPIDEMIC NEPHROPATHY (Infections and infestations) | 1 (1) | 0 (0)
EPIGLOTTITIS (Infections and infestations) | 2 (2) | 0 (0)
ERYSIPELAS (Infections and infestations) | 18 (19) | 14 (15)
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 1 (1) | 1 (1)
ESCHERICHIA INFECTION (Infections and infestations) | 1 (1) | 1 (1)
ESCHERICHIA SEPSIS (Infections and infestations) | 3 (3) | 2 (2)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
EYE ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
FUNGAEMIA (Infections and infestations) | 0 (0) | 1 (1)
GANGRENE (Infections and infestations) | 3 (3) | 1 (1)
GASTRIC INFECTION (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 37 (39) | 36 (37)
GASTROENTERITIS ESCHERICHIA COLI (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS NOROVIRUS (Infections and infestations) | 0 (0) | 1 (1)
GASTROENTERITIS VIRAL (Infections and infestations) | 4 (4) | 2 (2)
GASTROINTESTINAL BACTERIAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
GASTROINTESTINAL VIRAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
GINGIVAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
GRAFT INFECTION (Infections and infestations) | 3 (3) | 5 (5)
GROIN ABSCESS (Infections and infestations) | 7 (7) | 4 (4)
GROIN INFECTION (Infections and infestations) | 2 (2) | 0 (0)
H1N1 INFLUENZA (Infections and infestations) | 1 (1) | 3 (3)
HAEMATOMA INFECTION (Infections and infestations) | 1 (1) | 1 (1)
HELICOBACTER INFECTION (Infections and infestations) | 0 (0) | 1 (1)
HEPATITIS B (Infections and infestations) | 3 (3) | 0 (0)
HEPATITIS C (Infections and infestations) | 2 (2) | 1 (1)
HERPES SIMPLEX (Infections and infestations) | 1 (2) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 4 (4) | 3 (3)
HISTOPLASMOSIS (Infections and infestations) | 0 (0) | 1 (1)
HIV INFECTION (Infections and infestations) | 1 (1) | 0 (0)
IMPLANT SITE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
INCISION SITE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
INFECTED BITES (Infections and infestations) | 1 (1) | 0 (0)
INFECTED DERMAL CYST (Infections and infestations) | 1 (1) | 0 (0)
INFECTED SKIN ULCER (Infections and infestations) | 9 (9) | 9 (9)
INFECTION (Infections and infestations) | 5 (5) | 7 (7)
INFECTIOUS PERITONITIS (Infections and infestations) | 3 (4) | 1 (1)
INFECTIOUS PLEURAL EFFUSION (Infections and infestations) | 0 (0) | 2 (2)
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 5 (5) | 0 (0)
INFLUENZA (Infections and infestations) | 4 (4) | 1 (1)
INFUSION SITE INFECTION (Infections and infestations) | 0 (0) | 1 (1)
LABYRINTHITIS (Infections and infestations) | 2 (2) | 4 (4)
LIVER ABSCESS (Infections and infestations) | 3 (3) | 1 (1)
LOBAR PNEUMONIA (Infections and infestations) | 20 (20) | 23 (23)
LOCALISED INFECTION (Infections and infestations) | 9 (9) | 6 (8)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 8 (9) | 6 (6)
LOWER RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 1 (1) | 0 (0)
LUNG ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
LUNG INFECTION (Infections and infestations) | 6 (6) | 3 (3)
LYME DISEASE (Infections and infestations) | 1 (1) | 0 (0)
LYMPHANGITIS (Infections and infestations) | 1 (1) | 0 (0)
MASTOIDITIS (Infections and infestations) | 0 (0) | 1 (1)
MEDIASTINITIS (Infections and infestations) | 2 (2) | 1 (1)
MENINGITIS (Infections and infestations) | 0 (0) | 1 (1)
MENINGITIS ASEPTIC (Infections and infestations) | 0 (0) | 1 (1)
MENINGITIS BACTERIAL (Infections and infestations) | 1 (1) | 0 (0)
MENINGITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0)
MYCOBACTERIUM AVIUM COMPLEX INFECTION (Infections and infestations) | 0 (0) | 1 (1)
NECROTISING FASCIITIS (Infections and infestations) | 1 (1) | 1 (1)
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 0 (0) | 2 (2)
ONYCHOMYCOSIS (Infections and infestations) | 1 (1) | 0 (0)
ORAL CANDIDIASIS (Infections and infestations) | 1 (1) | 0 (0)
ORAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
ORCHITIS (Infections and infestations) | 3 (3) | 4 (4)
OSTEOMYELITIS (Infections and infestations) | 17 (19) | 14 (16)
OSTEOMYELITIS CHRONIC (Infections and infestations) | 0 (0) | 2 (2)
OTITIS EXTERNA (Infections and infestations) | 1 (1) | 0 (0)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 1 (1)
OTITIS MEDIA CHRONIC (Infections and infestations) | 0 (0) | 1 (1)
PAROTITIS (Infections and infestations) | 1 (1) | 0 (0)
PERICARDITIS INFECTIVE (Infections and infestations) | 0 (0) | 1 (2)
PERIDIVERTICULAR ABSCESS (Infections and infestations) | 1 (1) | 1 (1)
PERINEAL ABSCESS (Infections and infestations) | 1 (1) | 1 (1)
PERINEPHRIC ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
PERIORBITAL CELLULITIS (Infections and infestations) | 1 (1) | 1 (1)
PERIRECTAL ABSCESS (Infections and infestations) | 2 (2) | 1 (1)
PERITONSILLAR ABSCESS (Infections and infestations) | 2 (2) | 0 (0)
PHARYNGITIS BACTERIAL (Infections and infestations) | 1 (1) | 0 (0)
PILONIDAL CYST (Infections and infestations) | 0 (0) | 1 (1)
PNEUMOCYSTIS JIROVECI PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 186 (205) | 167 (185)
PNEUMONIA BACTERIAL (Infections and infestations) | 3 (3) | 2 (2)
PNEUMONIA ESCHERICHIA (Infections and infestations) | 0 (0) | 1 (1)
PNEUMONIA FUNGAL (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA MYCOPLASMAL (Infections and infestations) | 0 (0) | 2 (2)
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 1 (1) | 2 (2)
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 2 (2) | 3 (3)
PNEUMONIA VIRAL (Infections and infestations) | 1 (1) | 1 (1)
POST PROCEDURAL CELLULITIS (Infections and infestations) | 0 (0) | 1 (1)
POST PROCEDURAL INFECTION (Infections and infestations) | 4 (4) | 4 (4)
POST PROCEDURAL SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
POSTOPERATIVE ABSCESS (Infections and infestations) | 2 (2) | 0 (0)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 21 (24) | 10 (10)
PSEUDOMEMBRANOUS COLITIS (Infections and infestations) | 0 (0) | 1 (1)
PSOAS ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
PULMONARY SEPSIS (Infections and infestations) | 12 (13) | 18 (18)
PULMONARY TUBERCULOSIS (Infections and infestations) | 2 (2) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 11 (11) | 10 (10)
PYELONEPHRITIS ACUTE (Infections and infestations) | 1 (1) | 3 (3)
RECTAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 8 (9) | 6 (6)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 (0) | 1 (1)
SALMONELLA SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
SALMONELLOSIS (Infections and infestations) | 1 (1) | 1 (1)
SCROTAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 34 (34) | 28 (29)
SEPTIC NECROSIS (Infections and infestations) | 1 (1) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 22 (22) | 13 (13)
SERRATIA INFECTION (Infections and infestations) | 1 (1) | 0 (0)
SIALOADENITIS (Infections and infestations) | 1 (1) | 0 (0)
SINUSITIS (Infections and infestations) | 3 (3) | 3 (3)
SINUSITIS BACTERIAL (Infections and infestations) | 0 (0) | 1 (1)
SKIN INFECTION (Infections and infestations) | 2 (2) | 1 (1)
SOFT TISSUE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
STAPHYLOCOCCAL ABSCESS (Infections and infestations) | 0 (0) | 1 (1)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 9 (9) | 4 (4)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1 (2) | 0 (0)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 4 (4) | 2 (2)
SUPERINFECTION (Infections and infestations) | 0 (0) | 1 (1)
SYPHILIS (Infections and infestations) | 1 (1) | 0 (0)
SYSTEMIC CANDIDA (Infections and infestations) | 1 (1) | 0 (0)
TONSILLITIS (Infections and infestations) | 1 (1) | 0 (0)
TOOTH ABSCESS (Infections and infestations) | 1 (1) | 2 (2)
TUBERCULOSIS (Infections and infestations) | 0 (0) | 1 (1)
TYPHUS (Infections and infestations) | 0 (0) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 9 (9) | 4 (4)
URINARY TRACT INFECTION (Infections and infestations) | 50 (53) | 62 (67)
URINARY TRACT INFECTION BACTERIAL (Infections and infestations) | 0 (0) | 1 (1)
URINARY TRACT INFECTION PSEUDOMONAL (Infections and infestations) | 0 (0) | 1 (1)
URINARY TRACT INFECTION STAPHYLOCOCCAL (Infections and infestations) | 0 (0) | 1 (1)
UROSEPSIS (Infections and infestations) | 10 (10) | 27 (27)
VAGINAL INFECTION (Infections and infestations) | 2 (2) | 0 (0)
VARICELLA (Infections and infestations) | 0 (0) | 1 (1)
VESTIBULAR NEURONITIS (Infections and infestations) | 1 (1) | 2 (2)
VIRAL INFECTION (Infections and infestations) | 8 (8) | 11 (11)
VIRAL LABYRINTHITIS (Infections and infestations) | 1 (1) | 1 (1)
VIRAL MYOCARDITIS (Infections and infestations) | 0 (0) | 2 (2)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
WOUND ABSCESS (Infections and infestations) | 1 (1) | 1 (1)
WOUND INFECTION (Infections and infestations) | 6 (6) | 11 (11)
WOUND INFECTION PSEUDOMONAS (Infections and infestations) | 1 (1) | 0 (0)
WOUND INFECTION STAPHYLOCOCCAL (Infections and infestations) | 1 (1) | 0 (0)
WOUND SEPSIS (Infections and infestations) | 2 (2) | 1 (1)
ABDOMINAL WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
ACCIDENT (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
ACETABULUM FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 8 (8) | 8 (8)
ANAEMIA POSTOPERATIVE (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
ANASTOMOTIC COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ANASTOMOTIC STENOSIS (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 15 (16) | 17 (18)
ARTERIAL INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ARTHROPOD STING (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
BRAIN CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
BURNS THIRD DEGREE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CARBON MONOXIDE POISONING (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
CARDIAC FUNCTION DISTURBANCE POSTOPERATIVE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CARTILAGE INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
CHEMICAL EYE INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CHEST INJURY (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
CONCUSSION (Injury, poisoning and procedural complications) | 7 (8) | 4 (4)
CONFUSION POSTOPERATIVE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CONTUSION (Injury, poisoning and procedural complications) | 11 (14) | 7 (7)
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
CYSTITIS RADIATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
EAR INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ELECTRIC SHOCK (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
EXCORIATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
EXTRADURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FACE INJURY (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
FACIAL BONES FRACTURE (Injury, poisoning and procedural complications) | 10 (10) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 10 (10) | 11 (11)
FEBRILE NONHAEMOLYTIC TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 6 (6) | 4 (4)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 22 (23) | 16 (16)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
FLAIL CHEST (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
FOREARM FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
FOREIGN BODY (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
GASTROINTESTINAL STOMA COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
GUN SHOT WOUND (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
HAND FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
HEAD INJURY (Injury, poisoning and procedural complications) | 3 (3) | 8 (8)
HEAT EXHAUSTION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HEAT STROKE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 19 (19) | 16 (16)
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 9 (9) | 9 (10)
INCISION SITE HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
INCISION SITE PAIN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 9 (9) | 7 (7)
INJURY (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
INTERVERTEBRAL DISC INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
JAW FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 9 (10) | 9 (9)
JOINT INJURY (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
LACERATION (Injury, poisoning and procedural complications) | 10 (11) | 6 (6)
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
LIMB INJURY (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
LIMB TRAUMATIC AMPUTATION (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 6 (6)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
MENISCUS LESION (Injury, poisoning and procedural complications) | 8 (8) | 4 (4)
MULTIPLE DRUG OVERDOSE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 3 (3) | 6 (7)
MUSCLE RUPTURE (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
NERVE INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OPEN FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OPEN WOUND (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OPERATIVE HAEMORRHAGE (Injury, poisoning and procedural complications) | 19 (20) | 23 (23)
OVERDOSE (Injury, poisoning and procedural complications) | 4 (4) | 7 (7)
PATELLA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
PELVIC FRACTURE (Injury, poisoning and procedural complications) | 5 (5) | 3 (3)
PERIPROSTHETIC FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POISONING (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
POST PROCEDURAL DISCHARGE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 23 (24) | 39 (40)
POSTOPERATIVE ADHESION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
POSTOPERATIVE FEVER (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
POSTOPERATIVE ILEUS (Injury, poisoning and procedural complications) | 2 (2) | 5 (6)
POSTOPERATIVE RESPIRATORY DISTRESS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POSTOPERATIVE THORACIC PROCEDURE COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
POSTPERICARDIOTOMY SYNDROME (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
PROCEDURAL HYPOTENSION (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
PUBIS FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
RADIATION ASSOCIATED PAIN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
RADIATION INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
RADIATION OESOPHAGITIS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
RIB FRACTURE (Injury, poisoning and procedural complications) | 7 (7) | 12 (12)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 16 (16) | 13 (13)
SCAPULA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SEROMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SKIN FLAP NECROSIS (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SKULL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SNAKE BITE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SOFT TISSUE INJURY (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
SPINAL COLUMN INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 5 (6)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 6 (6) | 2 (2)
SPLENIC RUPTURE (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
STAB WOUND (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
STERNAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
STRUCK BY LIGHTNING (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 11 (12) | 14 (14)
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 5 (5) | 11 (11)
THERMAL BURN (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 6 (6)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
TRANSFUSION-RELATED ACUTE LUNG INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
TRAUMATIC ARTHRITIS (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
TRAUMATIC HAEMATOMA (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
TRAUMATIC HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
TRAUMATIC INTRACRANIAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
TRAUMATIC LIVER INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
ULNA FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
VACCINATION COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
VASCULAR INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
WOUND (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 6 (6) | 0 (0)
WOUND EVISCERATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
WOUND HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
WOUND NECROSIS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2) | 2 (2)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1 (1) | 3 (3)
BLOOD GLUCOSE DECREASED (Investigations) | 1 (1) | 0 (0)
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 1 (1) | 0 (0)
CARDIAC STRESS TEST ABNORMAL (Investigations) | 1 (1) | 1 (1)
CLOSTRIDIUM TEST POSITIVE (Investigations) | 1 (1) | 0 (0)
EJECTION FRACTION (Investigations) | 1 (1) | 0 (0)
EJECTION FRACTION ABNORMAL (Investigations) | 0 (0) | 1 (1)
EJECTION FRACTION DECREASED (Investigations) | 0 (0) | 2 (2)
EXERCISE ELECTROCARDIOGRAM ABNORMAL (Investigations) | 0 (0) | 1 (1)
EXERCISE TEST ABNORMAL (Investigations) | 1 (1) | 0 (0)
HAEMATOCRIT DECREASED (Investigations) | 1 (1) | 0 (0)
HAEMOGLOBIN DECREASED (Investigations) | 1 (1) | 2 (2)
HEPATIC ENZYME ABNORMAL (Investigations) | 0 (0) | 1 (1)
HEPATIC ENZYME INCREASED (Investigations) | 0 (0) | 1 (1)
HIV TEST POSITIVE (Investigations) | 1 (1) | 0 (0)
INTERNATIONAL NORMALISED RATIO INCREASED (Investigations) | 2 (2) | 1 (1)
OCCULT BLOOD (Investigations) | 0 (0) | 1 (1)
OCCULT BLOOD POSITIVE (Investigations) | 3 (3) | 1 (1)
PLATELET COUNT ABNORMAL (Investigations) | 2 (2) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 7 (7) | 4 (4)
PRECANCEROUS CELLS PRESENT (Investigations) | 0 (0) | 1 (1)
PROTEIN URINE PRESENT (Investigations) | 1 (1) | 0 (0)
PULMONARY FUNCTION TEST DECREASED (Investigations) | 1 (1) | 0 (0)
RED BLOOD CELL COUNT DECREASED (Investigations) | 1 (1) | 0 (0)
RED BLOOD CELLS URINE POSITIVE (Investigations) | 1 (1) | 0 (0)
TRANSAMINASES INCREASED (Investigations) | 1 (1) | 0 (0)
WEIGHT DECREASED (Investigations) | 0 (0) | 1 (1)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 (1) | 0 (0)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 33 (34) | 28 (28)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 12 (12) | 22 (23)
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 12 (13) | 16 (17)
DIABETIC COMPLICATION (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
DIABETIC FOOT (Metabolism and nutrition disorders) | 3 (3) | 3 (4)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 5 (6) | 9 (10)
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 3 (3) | 4 (4)
FLUID OVERLOAD (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
GOUT (Metabolism and nutrition disorders) | 5 (5) | 10 (11)
HAEMOSIDEROSIS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 19 (19) | 18 (19)
HYPERKALAEMIA (Metabolism and nutrition disorders) | 10 (10) | 7 (7)
HYPERVOLAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 17 (18) | 23 (26)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 9 (9) | 6 (6)
HYPOPHAGIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
IRON METABOLISM DISORDER (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
MALNUTRITION (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
OBESITY (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
TYPE 1 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 5 (5) | 7 (7)
VITAMIN B12 DEFICIENCY (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (7)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 20 (23) | 16 (16)
ARTHROFIBROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 16 (18) | 11 (11)
BONE CYST (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BONE FISTULA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
BURSITIS (Musculoskeletal and connective tissue disorders) | 7 (7) | 2 (2)
CERVICAL SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4)
CHONDROMALACIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
COMPARTMENT SYNDROME (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4)
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
DUPUYTREN'S CONTRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
EXOSTOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
FIBROMYALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1)
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
FRACTURE NONUNION (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
GOUTY ARTHRITIS (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
HAEMARTHROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 7 (8) | 8 (8)
INTERVERTEBRAL DISC DISORDER (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 31 (31) | 19 (19)
LIGAMENT LAXITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 14 (14) | 7 (7)
MENISCAL DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MONARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCLE ATROPHY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCLE HAEMORRHAGE (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 27 (29) | 41 (44)
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 17 (17) | 15 (15)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 5 (6) | 2 (2)
MYOFASCIAL PAIN SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
MYOSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
NEUROPATHIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OSTEITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 84 (89) | 71 (76)
OSTEOCHONDROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
OSTEOLYSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (5)
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PERIARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
POLYARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
POLYMYALGIA RHEUMATICA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
PSEUDARTHROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 9 (9) | 14 (14)
SCOLIOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 21 (21) | 14 (14)
SPINAL DISORDER (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 12 (12) | 8 (8)
SPONDYLITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
SPONDYLOLISTHESIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
SYMPATHETIC POSTERIOR CERVICAL SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
TENDON DISORDER (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
TENDON NECROSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
TENOSYNOVITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
TRIGGER FINGER (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
VERTEBRAL WEDGING (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ACUTE LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
ACUTE LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
ADENOMA BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ADRENAL ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
ADRENAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
ANAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
ANAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ANOGENITAL WARTS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
ASTROCYTOMA MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ATYPICAL FIBROXANTHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 (20) | 14 (15)
BENIGN CARDIAC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BENIGN LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
BENIGN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
BENIGN NEOPLASM OF BLADDER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
BENIGN NEOPLASM OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BENIGN NEOPLASM OF TESTIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BENIGN NEOPLASM OF THYROID GLAND (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
BENIGN RENAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BENIGN SALIVARY GLAND NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
BILE DUCT CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 5 (5)
BILIARY CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
BILIARY NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 21 (21) | 25 (25)
BLADDER CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 5 (6)
BLADDER NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
BLADDER PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BLADDER TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
BONE NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BRAIN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19 (19) | 17 (17)
BREAST CANCER IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BREAST CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
BREAST CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
BREAST NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
BRONCHIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 4 (4)
BRONCHIOLOALVEOLAR CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
CARCINOID TUMOUR OF THE DUODENUM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CARCINOMA IN SITU (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CERVIX CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CERVIX CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
CHLOROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
CHOLESTEATOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
CHONDROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CHONDROSARCOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CHOROID MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CHRONIC LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 7 (7)
CHRONIC MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 1 (1)
COLON ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 3 (3)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 25 (25) | 27 (27)
COLON CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 9 (9)
COLON CANCER STAGE 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
COLON NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
COLORECTAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
CONNECTIVE TISSUE NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
ENDOMETRIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
ESSENTIAL THROMBOCYTHAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
FIBROUS HISTIOCYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
GASTRIC ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 6 (6)
GASTRIC CANCER STAGE III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
GASTRIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
GASTROINTESTINAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
GASTROINTESTINAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
GASTROINTESTINAL TRACT ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
GLIOBLASTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
GLIOBLASTOMA MULTIFORME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
HAEMANGIOMA OF SPLEEN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
HEPATIC ANGIOSARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
HEPATIC CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
HEPATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 6 (6)
HEPATIC NEOPLASM MALIGNANT RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
HODGKIN'S DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
HYPOPHARYNGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
HYPOPHARYNGEAL CANCER STAGE III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
INFECTED NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
INTESTINAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
INTRADUCTAL PAPILLOMA OF BREAST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
KERATOACANTHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LARGE CELL CARCINOMA OF THE RESPIRATORY TRACT STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LARGE CELL LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LARGE GRANULAR LYMPHOCYTOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LARYNGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
LARYNGEAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LARYNGEAL CANCER STAGE 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LARYNGEAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LEIOMYOSARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LEIOMYOSARCOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LIP AND/OR ORAL CAVITY CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LIP NEOPLASM MALIGNANT STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
LIPOSARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 12 (12)
LUNG ADENOCARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 4 (4)
LUNG ADENOCARCINOMA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 27 (27) | 18 (18)
LUNG CARCINOMA CELL TYPE UNSPECIFIED STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 29 (29) | 29 (29)
LUNG SQUAMOUS CELL CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LUNG SQUAMOUS CELL CARCINOMA STAGE I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LUNG SQUAMOUS CELL CARCINOMA STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LUNG SQUAMOUS CELL CARCINOMA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 4 (4)
LYMPHANGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
LYMPHOCYTIC LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 3 (3)
MALIGNANT FIBROUS HISTIOCYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
MALIGNANT GLIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 3 (3)
MALIGNANT NEOPLASM OF EYE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MANTLE CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
MELANOMA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MENINGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
MENINGIOMA BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MESOTHELIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
MESOTHELIOMA MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3)
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
METASTASES TO LIVER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
METASTASES TO LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
METASTASES TO PERITONEUM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
METASTASIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
METASTATIC BRONCHIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
METASTATIC CARCINOMA OF THE BLADDER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
METASTATIC GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 6 (6)
METASTATIC LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
METASTATIC MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 6 (6)
METASTATIC SALIVARY GLAND CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
METASTATIC SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
MONOCLONAL GAMMOPATHY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
MULTIPLE MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 3 (3)
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 1 (1)
MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
NASOPHARYNGEAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
NASOPHARYNGEAL CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
NEOPLASM PROSTATE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
NEUROENDOCRINE CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
NEUROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
NON-HODGKIN'S LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
NON-HODGKIN'S LYMPHOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
NON-HODGKIN'S LYMPHOMA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
NON-HODGKIN'S LYMPHOMA STAGE II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 5 (5)
NON-SMALL CELL LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
NON-SMALL CELL LUNG CANCER STAGE IIIB (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
NON-SMALL CELL LUNG CANCER STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OESOPHAGEAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
OESOPHAGEAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
OESOPHAGEAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 3 (3)
OESOPHAGEAL SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
ORAL CAVITY CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
ORAL PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OROPHARYNGEAL CANCER STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OSTEOCHONDROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OVARIAN ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OVARIAN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OVARIAN CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
OVARIAN EPITHELIAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OVARIAN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 7 (7)
PANCREATIC CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (9) | 10 (10)
PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PARAPROTEINAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PARATHYROID TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PENIS CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PENIS CARCINOMA STAGE II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PHARYNGEAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PITUITARY TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
PITUITARY TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
PLEURAL MESOTHELIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
POLYCYTHAEMIA VERA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 54 (54) | 38 (39)
PROSTATE CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 9 (9)
PROSTATE CANCER RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
PROSTATE CANCER STAGE I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PROSTATE CANCER STAGE II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
PROSTATE CANCER STAGE IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PROSTATIC ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
RECTAL ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 (13) | 4 (4)
RECTOSIGMOID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
RENAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 3 (3)
RENAL CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
RENAL CANCER STAGE III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 7 (7)
RENAL CELL CARCINOMA RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
RENAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
RENAL ONCOCYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
RHABDOMYOSARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SALIVARY GLAND CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SALIVARY GLAND NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
SEBORRHOEIC KERATOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SKIN CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
SKIN NEOPLASM BLEEDING (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SMALL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SMALL CELL LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
SMALL CELL LUNG CANCER STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 7 (7)
SMALL INTESTINE CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
SMALL INTESTINE CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 8 (8)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
SQUAMOUS CELL CARCINOMA OF THE CERVIX (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
T-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
THYMOMA MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
THYROID ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
THYROID CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
THYROID CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
TONGUE NEOPLASM MALIGNANT STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
TONSIL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 9 (10)
TRANSITIONAL CELL CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
URETERAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
URETERIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
UTERINE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 4 (4)
UTERINE NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
VULVAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
ALTERED STATE OF CONSCIOUSNESS (Nervous system disorders) | 1 (1) | 0 (0)
AMYOTROPHIC LATERAL SCLEROSIS (Nervous system disorders) | 1 (1) | 3 (3)
ATAXIA (Nervous system disorders) | 1 (1) | 0 (0)
AUTONOMIC NERVOUS SYSTEM IMBALANCE (Nervous system disorders) | 1 (1) | 0 (0)
BASAL GANGLIA HAEMORRHAGE (Nervous system disorders) | 1 (1) | 0 (0)
BRAIN OEDEMA (Nervous system disorders) | 0 (0) | 1 (1)
BRAIN STEM HAEMORRHAGE (Nervous system disorders) | 0 (0) | 2 (2)
CAROTID ARTERY ANEURYSM (Nervous system disorders) | 0 (0) | 1 (1)
CAROTID ARTERY STENOSIS (Nervous system disorders) | 1 (1) | 2 (2)
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 1 (1) | 1 (1)
CAUDA EQUINA SYNDROME (Nervous system disorders) | 1 (1) | 1 (1)
CEREBRAL AMYLOID ANGIOPATHY (Nervous system disorders) | 0 (0) | 1 (1)
CEREBRAL CYST (Nervous system disorders) | 0 (0) | 1 (1)
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 2 (2) | 6 (6)
CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 2 (2)
CEREBROVASCULAR INSUFFICIENCY (Nervous system disorders) | 1 (1) | 0 (0)
CERVICAL MYELOPATHY (Nervous system disorders) | 2 (2) | 3 (3)
CERVICOBRACHIAL SYNDROME (Nervous system disorders) | 1 (1) | 6 (6)
CNS VENTRICULITIS (Nervous system disorders) | 1 (1) | 0 (0)
COGNITIVE DISORDER (Nervous system disorders) | 1 (1) | 0 (0)
COMA (Nervous system disorders) | 1 (1) | 0 (0)
COMPLEX PARTIAL SEIZURES (Nervous system disorders) | 0 (0) | 2 (2)
COMPLEX REGIONAL PAIN SYNDROME (Nervous system disorders) | 0 (0) | 1 (1)
COMPLICATED MIGRAINE (Nervous system disorders) | 1 (1) | 2 (2)
CONVULSION (Nervous system disorders) | 24 (27) | 18 (19)
CRANIAL NERVE PARALYSIS (Nervous system disorders) | 0 (0) | 2 (2)
CUBITAL TUNNEL SYNDROME (Nervous system disorders) | 1 (1) | 0 (0)
DEMENTIA (Nervous system disorders) | 4 (4) | 4 (4)
DEMENTIA ALZHEIMER'S TYPE (Nervous system disorders) | 2 (2) | 1 (1)
DEMYELINATING POLYNEUROPATHY (Nervous system disorders) | 1 (2) | 0 (0)
DIABETIC COMA (Nervous system disorders) | 0 (0) | 1 (1)
DIABETIC NEUROPATHY (Nervous system disorders) | 2 (2) | 3 (3)
DIZZINESS (Nervous system disorders) | 6 (6) | 16 (16)
DIZZINESS EXERTIONAL (Nervous system disorders) | 1 (1) | 0 (0)
DIZZINESS POSTURAL (Nervous system disorders) | 1 (1) | 0 (0)
DYSAESTHESIA (Nervous system disorders) | 1 (1) | 0 (0)
DYSARTHRIA (Nervous system disorders) | 3 (3) | 1 (1)
ENCEPHALITIS (Nervous system disorders) | 1 (1) | 0 (0)
ENCEPHALOMYELITIS (Nervous system disorders) | 0 (0) | 1 (1)
ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 1 (1)
EPILEPSY (Nervous system disorders) | 15 (15) | 20 (22)
FACIAL PARESIS (Nervous system disorders) | 0 (0) | 1 (1)
GRAND MAL CONVULSION (Nervous system disorders) | 2 (2) | 3 (3)
GUILLAIN-BARRE SYNDROME (Nervous system disorders) | 1 (1) | 2 (2)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 42 (43) | 75 (75)
HAEMORRHAGIC CEREBRAL INFARCTION (Nervous system disorders) | 1 (1) | 1 (1)
HAEMORRHAGIC STROKE (Nervous system disorders) | 0 (0) | 2 (2)
HAEMORRHAGIC TRANSFORMATION STROKE (Nervous system disorders) | 1 (1) | 6 (6)
HEADACHE (Nervous system disorders) | 7 (7) | 9 (10)
HEMIANOPIA (Nervous system disorders) | 1 (1) | 0 (0)
HEMIPARESIS (Nervous system disorders) | 1 (1) | 4 (4)
HYDROCEPHALUS (Nervous system disorders) | 2 (2) | 1 (1)
HYPERTENSIVE ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 1 (1)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1)
HYPOGLYCAEMIC COMA (Nervous system disorders) | 1 (1) | 2 (2)
HYPOXIC-ISCHAEMIC ENCEPHALOPATHY (Nervous system disorders) | 4 (4) | 0 (0)
IIIRD NERVE PARALYSIS (Nervous system disorders) | 1 (1) | 1 (1)
INTERCOSTAL NEURALGIA (Nervous system disorders) | 1 (1) | 1 (1)
INTRACRANIAL ANEURYSM (Nervous system disorders) | 0 (0) | 3 (3)
INTRACRANIAL HAEMATOMA (Nervous system disorders) | 0 (0) | 1 (1)
INTRACRANIAL HYPOTENSION (Nervous system disorders) | 1 (1) | 0 (0)
INTRAVENTRICULAR HAEMORRHAGE (Nervous system disorders) | 0 (0) | 1 (1)
LETHARGY (Nervous system disorders) | 0 (0) | 1 (1)
LEUKOENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 1 (1)
LEWIS-SUMNER SYNDROME (Nervous system disorders) | 0 (0) | 1 (1)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 (1) | 3 (3)
LUMBAR RADICULOPATHY (Nervous system disorders) | 4 (4) | 2 (2)
MENTAL IMPAIRMENT (Nervous system disorders) | 0 (0) | 1 (1)
METABOLIC ENCEPHALOPATHY (Nervous system disorders) | 3 (3) | 0 (0)
MIGRAINE (Nervous system disorders) | 8 (8) | 6 (7)
MONOPLEGIA (Nervous system disorders) | 1 (1) | 0 (0)
MYELOPATHY (Nervous system disorders) | 1 (1) | 0 (0)
MYOCLONUS (Nervous system disorders) | 1 (1) | 0 (0)
NERVE COMPRESSION (Nervous system disorders) | 1 (1) | 2 (2)
NERVE ROOT COMPRESSION (Nervous system disorders) | 0 (0) | 1 (1)
NERVOUS SYSTEM DISORDER (Nervous system disorders) | 0 (0) | 1 (1)
NEURALGIA (Nervous system disorders) | 0 (0) | 1 (1)
NEURITIS (Nervous system disorders) | 2 (2) | 0 (0)
NEUROLOGICAL SYMPTOM (Nervous system disorders) | 0 (0) | 1 (1)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 (1) | 1 (1)
NORMAL PRESSURE HYDROCEPHALUS (Nervous system disorders) | 0 (0) | 3 (3)
PARAESTHESIA (Nervous system disorders) | 1 (1) | 5 (5)
PARAPARESIS (Nervous system disorders) | 0 (0) | 1 (1)
PARAPLEGIA (Nervous system disorders) | 1 (1) | 0 (0)
PARKINSON'S DISEASE (Nervous system disorders) | 4 (5) | 5 (6)
PARKINSONISM (Nervous system disorders) | 0 (0) | 1 (1)
PARTIAL SEIZURES (Nervous system disorders) | 2 (2) | 1 (1)
PARTIAL SEIZURES WITH SECONDARY GENERALISATION (Nervous system disorders) | 1 (1) | 0 (0)
PERIPHERAL NERVE LESION (Nervous system disorders) | 1 (1) | 0 (0)
POLYNEUROPATHY (Nervous system disorders) | 1 (1) | 4 (5)
PRESYNCOPE (Nervous system disorders) | 20 (20) | 21 (22)
PUTAMEN HAEMORRHAGE (Nervous system disorders) | 0 (0) | 1 (1)
QUADRIPARESIS (Nervous system disorders) | 1 (1) | 0 (0)
RADICULITIS (Nervous system disorders) | 0 (0) | 2 (2)
RADICULOPATHY (Nervous system disorders) | 2 (2) | 1 (1)
SCIATICA (Nervous system disorders) | 7 (8) | 2 (2)
SEDATION (Nervous system disorders) | 1 (1) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 1 (1) | 0 (0)
SPINAL CLAUDICATION (Nervous system disorders) | 0 (0) | 2 (2)
SPINAL CORD COMPRESSION (Nervous system disorders) | 1 (1) | 0 (0)
STATUS EPILEPTICUS (Nervous system disorders) | 1 (1) | 2 (2)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 3 (3) | 5 (5)
SYNCOPE (Nervous system disorders) | 60 (65) | 81 (87)
SYRINGOMYELIA (Nervous system disorders) | 0 (0) | 1 (1)
TENSION HEADACHE (Nervous system disorders) | 1 (1) | 0 (0)
THORACIC OUTLET SYNDROME (Nervous system disorders) | 0 (0) | 1 (1)
TRANSIENT GLOBAL AMNESIA (Nervous system disorders) | 2 (2) | 2 (2)
TREMOR (Nervous system disorders) | 0 (0) | 1 (1)
TRIGEMINAL NEURALGIA (Nervous system disorders) | 0 (0) | 2 (2)
ULNAR NEURITIS (Nervous system disorders) | 1 (1) | 0 (0)
UPPER MOTOR NEURONE LESION (Nervous system disorders) | 0 (0) | 1 (2)
VASCULAR DEMENTIA (Nervous system disorders) | 0 (0) | 2 (3)
VASCULAR PARKINSONISM (Nervous system disorders) | 1 (1) | 0 (0)
VERTEBRAL ARTERY STENOSIS (Nervous system disorders) | 0 (0) | 1 (1)
VIITH NERVE PARALYSIS (Nervous system disorders) | 4 (4) | 2 (2)
VITH NERVE PARALYSIS (Nervous system disorders) | 0 (0) | 2 (2)
VOCAL CORD PARALYSIS (Nervous system disorders) | 0 (0) | 1 (1)
WERNICKE'S ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 1 (1)
ABORTION MISSED (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
ADJUSTMENT DISORDER (Psychiatric disorders) | 0 (0) | 1 (1)
ALCOHOL ABUSE (Psychiatric disorders) | 2 (2) | 1 (1)
ALCOHOLISM (Psychiatric disorders) | 2 (4) | 2 (2)
ANXIETY (Psychiatric disorders) | 9 (9) | 10 (10)
ANXIETY DISORDER (Psychiatric disorders) | 1 (1) | 0 (0)
BIPOLAR DISORDER (Psychiatric disorders) | 2 (2) | 2 (2)
BIPOLAR I DISORDER (Psychiatric disorders) | 0 (0) | 2 (2)
COMPLETED SUICIDE (Psychiatric disorders) | 3 (3) | 6 (6)
CONFUSIONAL STATE (Psychiatric disorders) | 5 (5) | 7 (7)
CONVERSION DISORDER (Psychiatric disorders) | 1 (1) | 0 (0)
DELIRIUM (Psychiatric disorders) | 4 (4) | 2 (2)
DEPRESSED MOOD (Psychiatric disorders) | 0 (0) | 2 (2)
DEPRESSION (Psychiatric disorders) | 19 (20) | 18 (19)
HALLUCINATION (Psychiatric disorders) | 0 (0) | 2 (2)
MAJOR DEPRESSION (Psychiatric disorders) | 4 (4) | 8 (8)
MANIA (Psychiatric disorders) | 1 (1) | 0 (0)
MENTAL DISORDER (Psychiatric disorders) | 1 (1) | 1 (1)
MENTAL STATUS CHANGES (Psychiatric disorders) | 2 (2) | 4 (4)
PANIC ATTACK (Psychiatric disorders) | 2 (2) | 1 (1)
POLYDIPSIA PSYCHOGENIC (Psychiatric disorders) | 1 (1) | 0 (0)
POST STROKE DEPRESSION (Psychiatric disorders) | 0 (0) | 3 (3)
PSYCHOTIC DISORDER (Psychiatric disorders) | 3 (3) | 1 (1)
RESTLESSNESS (Psychiatric disorders) | 0 (0) | 1 (1)
SCHIZOPHRENIA (Psychiatric disorders) | 1 (1) | 0 (0)
SOMATOFORM DISORDER (Psychiatric disorders) | 1 (2) | 1 (1)
STRESS (Psychiatric disorders) | 0 (0) | 1 (1)
SUBSTANCE ABUSE (Psychiatric disorders) | 0 (0) | 1 (1)
SUICIDAL IDEATION (Psychiatric disorders) | 6 (7) | 5 (5)
SUICIDE ATTEMPT (Psychiatric disorders) | 11 (11) | 7 (7)
TRANSIENT PSYCHOSIS (Psychiatric disorders) | 1 (1) | 1 (1)
ACUTE PRERENAL FAILURE (Renal and urinary disorders) | 2 (2) | 1 (1)
AZOTAEMIA (Renal and urinary disorders) | 1 (1) | 0 (0)
BLADDER DISORDER (Renal and urinary disorders) | 1 (1) | 0 (0)
BLADDER NECK OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 2 (2)
BLADDER NECK SCLEROSIS (Renal and urinary disorders) | 1 (1) | 1 (1)
BLADDER OUTLET OBSTRUCTION (Renal and urinary disorders) | 1 (1) | 0 (0)
BLADDER PERFORATION (Renal and urinary disorders) | 0 (0) | 1 (1)
BLADDER PROLAPSE (Renal and urinary disorders) | 1 (1) | 1 (1)
BLADDER SPASM (Renal and urinary disorders) | 1 (1) | 0 (0)
BLADDER STENOSIS (Renal and urinary disorders) | 1 (3) | 0 (0)
CALCULUS BLADDER (Renal and urinary disorders) | 2 (2) | 3 (3)
CALCULUS URETERIC (Renal and urinary disorders) | 6 (6) | 6 (6)
CALCULUS URETHRAL (Renal and urinary disorders) | 2 (2) | 0 (0)
CALCULUS URINARY (Renal and urinary disorders) | 2 (2) | 3 (3)
CYSTITIS HAEMORRHAGIC (Renal and urinary disorders) | 0 (0) | 1 (1)
CYSTITIS NONINFECTIVE (Renal and urinary disorders) | 0 (0) | 1 (1)
DIABETIC NEPHROPATHY (Renal and urinary disorders) | 3 (3) | 1 (1)
DYSURIA (Renal and urinary disorders) | 1 (1) | 0 (0)
GLOMERULONEPHRITIS (Renal and urinary disorders) | 0 (0) | 1 (1)
GLOMERULONEPHRITIS MEMBRANOUS (Renal and urinary disorders) | 1 (1) | 0 (0)
HAEMATURIA (Renal and urinary disorders) | 38 (42) | 66 (72)
HAEMORRHAGE URINARY TRACT (Renal and urinary disorders) | 1 (1) | 5 (6)
HYDRONEPHROSIS (Renal and urinary disorders) | 0 (0) | 3 (3)
HYDROURETER (Renal and urinary disorders) | 1 (1) | 0 (0)
KIDNEY FIBROSIS (Renal and urinary disorders) | 0 (0) | 1 (1)
MICTURITION URGENCY (Renal and urinary disorders) | 1 (1) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 28 (33) | 22 (22)
NEPHROPATHY (Renal and urinary disorders) | 0 (0) | 3 (3)
NEPHROTIC SYNDROME (Renal and urinary disorders) | 2 (2) | 1 (1)
OBSTRUCTIVE UROPATHY (Renal and urinary disorders) | 1 (1) | 1 (1)
PELVI-URETERIC OBSTRUCTION (Renal and urinary disorders) | 1 (1) | 0 (0)
POLYURIA (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL ARTERY OCCLUSION (Renal and urinary disorders) | 1 (1) | 0 (0)
RENAL ARTERY STENOSIS (Renal and urinary disorders) | 1 (1) | 2 (2)
RENAL COLIC (Renal and urinary disorders) | 3 (3) | 3 (3)
RENAL CYST (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 40 (42) | 33 (34)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 54 (61) | 43 (44)
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 18 (18) | 9 (13)
RENAL IMPAIRMENT (Renal and urinary disorders) | 4 (4) | 3 (3)
RENAL INFARCT (Renal and urinary disorders) | 0 (0) | 1 (1)
RENAL MASS (Renal and urinary disorders) | 1 (1) | 2 (2)
RENAL TUBULAR NECROSIS (Renal and urinary disorders) | 1 (1) | 1 (1)
STAG HORN CALCULUS (Renal and urinary disorders) | 0 (0) | 1 (1)
STRESS URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 1 (1)
TUBULOINTERSTITIAL NEPHRITIS (Renal and urinary disorders) | 1 (1) | 0 (0)
URETERIC RUPTURE (Renal and urinary disorders) | 1 (1) | 0 (0)
URETERIC STENOSIS (Renal and urinary disorders) | 2 (3) | 0 (0)
URETHRAL OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 1 (1)
URETHRAL STENOSIS (Renal and urinary disorders) | 2 (2) | 5 (6)
URINARY BLADDER POLYP (Renal and urinary disorders) | 1 (1) | 1 (1)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 1 (1)
URINARY RETENTION (Renal and urinary disorders) | 14 (14) | 4 (4)
URINARY TRACT DISORDER (Renal and urinary disorders) | 1 (1) | 1 (1)
VESICOURETERIC REFLUX (Renal and urinary disorders) | 0 (0) | 1 (1)
BALANITIS (Reproductive system and breast disorders) | 1 (1) | 0 (0)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 27 (28) | 35 (36)
BREAST ENLARGEMENT (Reproductive system and breast disorders) | 0 (0) | 1 (1)
CYSTOCELE (Reproductive system and breast disorders) | 5 (5) | 0 (0)
ENDOMETRIAL HYPERPLASIA (Reproductive system and breast disorders) | 1 (1) | 2 (2)
EPIDIDYMITIS (Reproductive system and breast disorders) | 2 (2) | 0 (0)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 0 (0) | 1 (1)
FIBROCYSTIC BREAST DISEASE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
GENITAL HAEMORRHAGE (Reproductive system and breast disorders) | 2 (2) | 2 (2)
GENITAL TRACT INFLAMMATION (Reproductive system and breast disorders) | 1 (1) | 0 (0)
MENOMETRORRHAGIA (Reproductive system and breast disorders) | 0 (0) | 2 (2)
MENORRHAGIA (Reproductive system and breast disorders) | 2 (2) | 5 (6)
MENSTRUAL DISORDER (Reproductive system and breast disorders) | 0 (0) | 2 (2)
METRORRHAGIA (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ORCHITIS NONINFECTIVE (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OVARIAN CYST (Reproductive system and breast disorders) | 4 (4) | 3 (3)
PELVIC HAEMATOMA (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PELVIC PROLAPSE (Reproductive system and breast disorders) | 1 (1) | 0 (0)
POSTMENOPAUSAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PROSTATIC HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
PROSTATISM (Reproductive system and breast disorders) | 1 (1) | 1 (1)
PROSTATITIS (Reproductive system and breast disorders) | 4 (4) | 3 (3)
PROSTATOMEGALY (Reproductive system and breast disorders) | 1 (1) | 2 (2)
RECTOCELE (Reproductive system and breast disorders) | 1 (1) | 2 (2)
SPERMATOCELE (Reproductive system and breast disorders) | 1 (1) | 0 (0)
TESTICULAR OEDEMA (Reproductive system and breast disorders) | 1 (1) | 0 (0)
UTERINE CYST (Reproductive system and breast disorders) | 0 (0) | 1 (1)
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
UTERINE PROLAPSE (Reproductive system and breast disorders) | 2 (2) | 3 (3)
UTEROVAGINAL PROLAPSE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 1 (1)
VAGINAL LACERATION (Reproductive system and breast disorders) | 0 (0) | 1 (1)
VAGINAL PROLAPSE (Reproductive system and breast disorders) | 3 (3) | 0 (0)
VAGINAL ULCERATION (Reproductive system and breast disorders) | 0 (0) | 1 (1)
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 18 (19) | 7 (9)
ADENOIDAL DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
APNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
ASPHYXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 8 (13) | 12 (15)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
BRAIN HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
BRONCHIAL HYPERREACTIVITY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 75 (100) | 79 (112)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
DIAPHRAGMATIC PARALYSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 13 (13)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
DYSPNOEA PAROXYSMAL NOCTURNAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
EOSINOPHILIC PNEUMONIA ACUTE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 29 (30)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 13 (13)
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 7 (7)
HYDROTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HYPERVENTILATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HYPOVENTILATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
IDIOPATHIC PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
LARYNGEAL MASS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
LARYNGEAL STENOSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
LUNG CONSOLIDATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
NASAL POLYPS (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
NASAL SEPTUM DEVIATION (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
NASAL SEPTUM DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
NASAL TURBINATE HYPERTROPHY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OBSTRUCTIVE AIRWAYS DISORDER (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
PHARYNGEAL HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 13 (14)
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 12 (15) | 4 (4)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 9 (13)
PULMONARY CALCIFICATION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 45 (45) | 23 (24)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
PULMONARY INFARCTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY NECROSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 8 (8)
RESPIRATORY ACIDOSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 21 (22)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
SINUS POLYP (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6)
TONSILLAR HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
VOCAL CORD ATROPHY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
VOCAL CORD POLYP (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ANGIODERMATITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 6 (6) | 7 (7)
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
DERMATITIS (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
DERMATITIS EXFOLIATIVE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DERMATOMYOSITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
DIABETIC DERMOPATHY (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DIABETIC ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
DRY GANGRENE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
LEUKOCYTOCLASTIC VASCULITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
PEMPHIGOID (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PEMPHIGUS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PETECHIAE (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PSORIASIS (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
PURPURA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
SCAR (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SEGMENTED HYALINISING VASCULITIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
SKIN HAEMORRHAGE (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
SKIN NECROSIS (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 4 (4) | 7 (7)
STASIS DERMATITIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
SOCIAL PROBLEM (Social circumstances) | 0 (0) | 1 (1)
ABDOMINAL OPERATION (Surgical and medical procedures) | 0 (0) | 1 (1)
FINGER AMPUTATION (Surgical and medical procedures) | 1 (1) | 0 (0)
GASTRIC BANDING (Surgical and medical procedures) | 0 (0) | 1 (1)
HIP ARTHROPLASTY (Surgical and medical procedures) | 0 (0) | 1 (1)
INGUINAL HERNIA REPAIR (Surgical and medical procedures) | 1 (1) | 0 (0)
POLYPECTOMY (Surgical and medical procedures) | 0 (0) | 1 (1)
SPINAL DECOMPRESSION (Surgical and medical procedures) | 1 (1) | 0 (0)
SURGERY (Surgical and medical procedures) | 1 (1) | 0 (0)
ACCELERATED HYPERTENSION (Vascular disorders) | 2 (2) | 1 (1)
ANEURYSM (Vascular disorders) | 1 (1) | 0 (0)
ANEURYSM RUPTURED (Vascular disorders) | 0 (0) | 1 (1)
ANGIODYSPLASIA (Vascular disorders) | 1 (1) | 1 (1)
AORTIC ANEURYSM (Vascular disorders) | 18 (18) | 18 (18)
AORTIC ANEURYSM RUPTURE (Vascular disorders) | 8 (8) | 3 (5)
AORTIC DILATATION (Vascular disorders) | 0 (0) | 1 (1)
AORTIC DISSECTION (Vascular disorders) | 0 (0) | 1 (2)
AORTIC STENOSIS (Vascular disorders) | 3 (3) | 7 (7)
ARTERIAL DISORDER (Vascular disorders) | 0 (0) | 1 (1)
ARTERIAL HAEMORRHAGE (Vascular disorders) | 0 (0) | 1 (1)
ARTERIAL RUPTURE (Vascular disorders) | 0 (0) | 1 (2)
ARTERIOSCLEROSIS (Vascular disorders) | 1 (1) | 0 (0)
ARTERIOVENOUS FISTULA (Vascular disorders) | 1 (1) | 2 (2)
BLEEDING VARICOSE VEIN (Vascular disorders) | 1 (1) | 2 (3)
CIRCULATORY COLLAPSE (Vascular disorders) | 1 (1) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 22 (23) | 19 (20)
ESSENTIAL HYPERTENSION (Vascular disorders) | 0 (0) | 2 (2)
EXTREMITY NECROSIS (Vascular disorders) | 1 (1) | 1 (1)
FEMORAL ARTERY ANEURYSM (Vascular disorders) | 0 (0) | 1 (1)
HAEMATOMA (Vascular disorders) | 16 (17) | 25 (26)
HAEMODYNAMIC INSTABILITY (Vascular disorders) | 1 (1) | 1 (1)
HAEMORRHAGE (Vascular disorders) | 23 (24) | 36 (40)
HYPERTENSION (Vascular disorders) | 26 (26) | 27 (32)
HYPERTENSIVE CRISIS (Vascular disorders) | 31 (35) | 20 (25)
HYPERTENSIVE EMERGENCY (Vascular disorders) | 4 (4) | 4 (5)
HYPOPERFUSION (Vascular disorders) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 29 (29) | 31 (31)
HYPOVOLAEMIC SHOCK (Vascular disorders) | 1 (1) | 2 (2)
INTRA-ABDOMINAL HAEMORRHAGE (Vascular disorders) | 1 (1) | 0 (0)
LABILE BLOOD PRESSURE (Vascular disorders) | 1 (1) | 0 (0)
LYMPHATIC FISTULA (Vascular disorders) | 1 (1) | 0 (0)
LYMPHOCELE (Vascular disorders) | 1 (1) | 1 (1)
LYMPHOEDEMA (Vascular disorders) | 1 (1) | 0 (0)
MALIGNANT HYPERTENSION (Vascular disorders) | 2 (2) | 1 (1)
ORTHOSTATIC HYPERTENSION (Vascular disorders) | 1 (1) | 1 (1)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 20 (20) | 13 (15)
PERIPHERAL ARTERY ANEURYSM (Vascular disorders) | 1 (1) | 1 (1)
PERIPHERAL EMBOLISM (Vascular disorders) | 1 (1) | 0 (0)
PHLEBITIS (Vascular disorders) | 1 (1) | 0 (0)
POOR PERIPHERAL CIRCULATION (Vascular disorders) | 1 (1) | 0 (0)
RAYNAUD'S PHENOMENON (Vascular disorders) | 0 (0) | 1 (1)
SHOCK (Vascular disorders) | 1 (1) | 0 (0)
SUBCLAVIAN VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
TEMPORAL ARTERITIS (Vascular disorders) | 2 (2) | 1 (1)
VARICOSE VEIN (Vascular disorders) | 2 (2) | 3 (3)
VENOUS INSUFFICIENCY (Vascular disorders) | 0 (0) | 1 (1)
VENOUS THROMBOSIS (Vascular disorders) | 2 (2) | 2 (2)
WEGENER'S GRANULOMATOSIS (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=13166) | Vorapaxar (N=13186)
CHEST PAIN (General disorders) | 687 (785) | 672 (789)
DIZZINESS (Nervous system disorders) | 704 (781) | 662 (746)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 401 (513) | 807 (1044)
HYPERTENSION (Vascular disorders) | 736 (789) | 712 (761)

LIMITATIONS AND CAVEATS:
Prior to the completion of the study, based on a communication from the Data and Safety Monitoring Board, all participants who had experienced a stroke either before or during the study had study drug discontinued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigators agreed not to publish or publicly present any interim results of the study without the prior written consent of the sponsor. The investigator further agreed to provide to the sponsor review copies of abstracts or manuscripts for publication 45 days prior to submission.